CLINICAL TRIAL: NCT03473223
Title: A Phase 3, Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Investigate the Efficacy and Safety of CSL112 in Subjects With Acute Coronary Syndrome
Brief Title: Study to Investigate CSL112 in Subjects With Acute Coronary Syndrome
Acronym: AEGIS-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSL112_3001; 2017-000996-98 (EudraCT Number)
Record Dates: First submitted 2018-03-14; First posted 2018-03-22 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Acute Coronary Syndrome
Keywords: Coronary Artery Disease; Heart Disease; Cardiovascular Disease; Acute Myocardial Infarction; Heart Failure; Major adverse cardiovascular event; Multivessel disease; Peripheral artery disease; Cerebrovascular accident; Ischemic stroke; Hemorrhagic stroke; Atherosclerosis; Congestive heart failure; Valvular heart disease; Atrial Fibrillation; Hypertension
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease; Heart Diseases; Cardiovascular Diseases; Heart Failure; Peripheral Arterial Disease; Stroke; Ischemic Stroke; Hemorrhagic Stroke; Atherosclerosis; Heart Valve Diseases; Atrial Fibrillation; Hypertension | interventions — Apolipoprotein A-I; CSL112

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CSL112 (Experimental): Apolipoprotein A-I [human]
  Interventions: Biological: Apolipoprotein A-I [human] (apoA-I)
- Placebo (Placebo Comparator): 25% albumin solution diluted to 4.4%
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Apolipoprotein A-I [human] (apoA-I) — Apolipoprotein A-I [human] (apoA-I) purified from human plasma for intravenous administration
  Other Names: CSL112
  Arms: CSL112
Other: Placebo — 25% albumin solution diluted to 4.4%
  Arms: Placebo

SUMMARY:
This is a phase 3, multicenter, double-blind, randomized, placebo-controlled, parallel-group study to evaluate the efficacy and safety of CSL112 on reducing the risk of major adverse CV events [MACE - cardiovascular (CV) death, myocardial infarction (MI), and stroke] in subjects with acute coronary syndrome (ACS) diagnosed with either ST-segment elevation myocardial infarction (STEMI) or non-ST-segment elevation myocardial infarction (NSTEMI), including those managed with percutaneous coronary intervention (PCI) or medically managed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female least 18 years of age
* Evidence of myocardial necrosis, consistent with type I (spontaneous) MI
* No suspicion of acute kidney injury
* Evidence of multivessel coronary artery disease
* Presence of established cardiovascular risk factor(s):

  1. Diabetes mellitus on pharmacotherapy OR
  2. 2 or more of the following: age ≥ 65 years, prior history of MI, peripheral arterial disease

Exclusion Criteria:

* Ongoing hemodynamic instability
* Evidence of hepatobiliary disease
* Evidence of severe chronic kidney disease
* Plan to undergo scheduled coronary artery bypass graft surgery as treatment for the index MI
* Known history of allergies, hypersensitivity, or deficiencies to soy bean, peanut or albumin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18226 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Duffy, MD, Study Director — CSL Behring - Executive Director, Clinical Development - CV & Metabolism
Locations (903):
- United States (202):
  - 8400896 - Advanced Cardiovascular LLC, Alexander City, Alabama
  - 8400350 - Cardiology, PC, Birmingham, Alabama
  - 8400337 - Heart Center Research, LLC, Huntsville, Alabama
  - 8400713 - University of South Alabama College of Medicine, Mobile, Alabama
  - 8400556 - Mercy Gilbert Medical Center, Gilbert, Arizona
  - 8400747 - Phoenix V.A. Health Care System, Phoenix, Arizona
  - 8400772 - Mayo Clinic Arizona, Phoenix, Arizona
  - 8400996 - Southern Arizona V.A. Healthcare System, Tucson, Arizona
  - 8400645 - NEA Baptist Clinic, Jonesboro, Arkansas
  - 8400975 - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - 8401054 - Central Cardiology Medical Center, Bakersfield, California
  - 8400379 - John Muir Health and Cardiovascular Institute, Concord, California
  - 8400931 - Valley Clinical Trials, Covina, California
  - 8401103 - Orange Coast Memorial Hospital, Fountain Valley, California
  - 8401166 - Sharp Grossmont Hospital, La Mesa, California
  - 8401192 - South Orange County Surgical Medical Group, Laguna Hills, California
  - 8400596 - Long Beach Memorial Medical Center, Long Beach, California
  - 8400910 - Cardiovascular Innovation and Research Center, Long Beach, California
  - 8400597 - Los Alamitos Cardiovascular, Los Alamitos, California
  - 8400693 - University of California Los Angeles, Los Angeles, California
  - 8400717 - V.A. Greater Los Angeles Healthcare System, Los Angeles, California
  - 8400888 - Saint Jude Heritage Healthcare, Mission Viejo, California
  - 8400745 - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - 8400658 - Valley Clinical Trials, Inc., Northridge, California
  - 8400720 - Valley Clinical Trials, Pasadena, California
  - 8400787 - Riverside Community Hospital, Riverside, California
  - 8400694 - University of California San Diego Medical Center, San Diego, California
  - 8400703 - San Diego Cardiac Center, San Diego, California
  - 8400719 - V.A. San Diego Health Care System, San Diego, California
  - 8400909 - Ventura Clinical Trials, Ventura, California
  - 8400891 - John Muir Medical Center Walnu, Walnut Creek, California
  - 8400893 - Interventional Cardiology Medical Group, West Hills, California
  - 8400574 - Aurora Denver Cardiology Associates, Aurora, Colorado
  - 8400684 - UCHealth Memorial Hospital Central - Colorado Springs, Colorado Springs, Colorado
  - 8400997 - CardioVascular Institute of North Colorado Cardiology Clinic, Greeley, Colorado
  - 8400670 - Medical Center of the Rockies, Loveland, Colorado
  - 8400371 - Danbury Hospital, Danbury, Connecticut
  - 8401134 - Christiana Hospital, Newark, Delaware
  - 8400779 - MedStar Clinical Research Center, Washington D.C., District of Columbia
  - 8400688 - George Washington University Medical Center, Washington D.C., District of Columbia
  - 8400484 - Clearwater Cardiovascular and Interventional Consultants, Clearwater, Florida
  - 8400544 - Cardiology Research Associates, Daytona Beach, Florida
  - 8400930 - Lake Internal Medicine Assoc., Eustis, Florida
  - 8400613 - Jim Moran Heart and Vascular Center, Fort Lauderdale, Florida
  - 8401010 - Integrative Research Associates Inc., Fort Lauderdale, Florida
  - 8400490 - University of Florida, Gainesville, Florida
  - 8400517 - Shands Jacksonville Medical Center, Jacksonville, Florida
  - 8400985 - Optimus U Corp., Miami, Florida
  - 8400543 - Cardiology Partners Research Institute, Palm Beach Gardens, Florida
  - 8400542 - Cardiology Consultants, Pensacola, Florida
  - 8400557 - Clearwater Cardiovascular and Interventional Consultants, Safety Harbor, Florida
  - 8400686 - Intercoastal Medical Group, Sarasota, Florida
  - 8400736 - Pepin Heart Institute, Tampa, Florida
  - 8401011 - Cardiology Partners Research Institute, Wellington, Florida
  - 8401185 - Piedmont Heart Institute, Athens, Georgia
  - 8400376 - Emory University, Atlanta, Georgia
  - 8400918 - Augusta University, Augusta, Georgia
  - 8400849 - IACT Health, Columbus, Georgia
  - 8400655 - Atlanta V.A. Medical Center, Decatur, Georgia
  - 8401120 - Northeast Georgia Medical Center, Gainesville, Georgia
  - 8401157 - Memorial Health University Medical Center, Savannah, Georgia
  - 8400357 - Saint Luke's Boise Medical Center, Boise, Idaho
  - 8400610 - Jesse Brown V.A. Medical Center, Chicago, Illinois
  - 8401093 - Advanced Heart Care Group, Fairview Heights, Illinois
  - 8401000 - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - 8400785 - OSF Multi-Specialty Group, Peoria, Illinois
  - 8400361 - Midwest Cardiovascular Research, Elkhart, Indiana
  - 8400961 - Indiana Heart Physicians, Inc., Indianapolis, Indiana
  - 8400989 - Indiana Heart Hospital, Indianapolis, Indiana
  - 8400507 - The Saint Vincent Heart Center of Indiana, Indianapolis, Indiana
  - 8400576 - IU Health Ball Memorial Hospital Physicians, Inc, Muncie, Indiana
  - 8400882 - Reid Health, Richmond, Indiana
  - 8400618 - McFarland Clinic, PC, Ames, Iowa
  - 8400904 - Northeast Iowa Medical Education Foundation, Waterloo, Iowa
  - 8400678 - The Iowa Clinic, PC, West Des Moines, Iowa
  - 8400978 - Midwest Heart and Vascular, Overland Park, Kansas
  - 8400661 - Norton Cardiovascular Associates, Louisville, Kentucky
  - 8400368 - Cambridge Medical Trials, Alexandria, Louisiana
  - 8400862 - Cardiovascular Associates Research, Covington, Louisiana
  - 8401104 - Cardiovascular Institute of the South, Houma, Louisiana
  - 8400563 - Cardiovascular Institute of the South, Lafayette, Louisiana
  - 8401127 - Tulane University Health Science Center, New Orleans, Louisiana
  - 8401175 - Overton Brooks V.A. Medical Center, Shreveport, Louisiana
  - 8400483 - Eastern Maine Medical Center, Bangor, Maine
  - 8400812 - Maine Medical Center Bramhall Campus, Portland, Maine
  - 8401142 - Anne Arundel Health System, Annapolis, Maryland
  - 8401163 - Washington Adventist Hospital, Takoma Park, Maryland
  - 8400998 - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - 8400769 - Healthy Heart Cardiology, Grandville, Michigan
  - 8401141 - Western Michigan University Homer Striker MD School of Medicine, Kalamazoo, Michigan
  - 8400638 - Mid Michigan Regional Medical Center, Midland, Michigan
  - 8401092 - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - 8400861 - Ascension Providence Rochester Hospital, Rochester, Michigan
  - 8400372 - Covenant Medical Center, Saginaw, Michigan
  - 8400667 - Michigan Cardiovascular Institute, Saginaw, Michigan
  - 8401165 - Ascension Macomb-Oakland Hospital Warren Campus, Warren, Michigan
  - 8400625 - Michigan Heart and Vascular Institute, Ypsilanti, Michigan
  - 8400488 - Essentia Health, Duluth, Minnesota
  - 8400920 - Saint Lukes Hospital, Duluth, Minnesota
  - 8400364 - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - 8400752 - Regions Hospital, Saint Paul, Minnesota
  - 8400369 - HealthEast Saint Joseph's Hospital, Saint Paul, Minnesota
  - 8401168 - Jackson Heart Clinic, Jackson, Mississippi
  - 8400334 - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - 8401108 - University of Missouri Health System, Columbia, Missouri
  - 8400648 - Saint Luke's Cardiovascular Consultants, Kansas City, Missouri
  - 8400631 - North Kansas City Hospital, North Kansas City, Missouri
  - 8400622 - Mercy Medical Research Institute, Springfield, Missouri
  - 8400840 - Washington University, St Louis, Missouri
  - 8400091 - Glacier View Cardiology, Kalispell, Montana
  - 8400783 - Nebraska Heart Institute, Lincoln, Nebraska
  - 8400689 - University Medical Center, Las Vegas, Nevada
  - 8400545 - Advanced Heart Care LLC, Bridgewater, New Jersey
  - 8400835 - Cooper University Hospital, Camden, New Jersey
  - 8400836 - Our Lady of Lourdes Medical Center, Camden, New Jersey
  - 8401178 - Jersey Shore University Medical Center Meridian Health, Neptune City, New Jersey
  - 8401144 - Saint Michael's Medical Center, Newark, New Jersey
  - 8400572 - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - 8401189 - Cardiovascular Associates of the Delaware Valley, Vineland, New Jersey
  - 8400742 - VMG Cardiology, Westwood, Westwood, New Jersey
  - 8400360 - Buffalo Heart Group, Buffalo, New York
  - 8401028 - Buffalo V.A. Medical Center, Buffalo, New York
  - 8400677 - Saint Joseph's Hospital Cardiac Catheterization Associates, Liverpool, New York
  - 8400380 - Mount Sinai Medical Center, New York, New York
  - 8401119 - Lenox Hill Hospital, New York, New York
  - 8401154 - Rochester General Hospital, Rochester, New York
  - 8400847 - University of Rochester Medical Center-Strong Memorial Hospital, Rochester, New York
  - 8400626 - Montefiore Medical Center - Albert Einstein College of Medicine, The Bronx, New York
  - 8400636 - Jacobi Medical Center, The Bronx, New York
  - 8400726 - Westchester Medical Center, Valhalla, New York
  - 8401027 - UNC Hospitals Heart and Vascular Center at Meadowmont, Chapel Hill, North Carolina
  - 8400733 - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - 8400489 - Duke University Hospital, Durham, North Carolina
  - 8400491 - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - 8400366 - High Point Regional Hospital, High Point, North Carolina
  - 8400916 - Southeastern Cardiology & Cardiovascular Clinic, Lumberton, North Carolina
  - 8400887 - Matthews Medical Center, Matthews, North Carolina
  - 8400889 - NC Heart and Vascular Research, Raleigh, North Carolina
  - 8400322 - Wake Forest University Health Sciences, Dept. of Cardiovascular Medicine, Winston-Salem, North Carolina
  - 8400651 - Sanford Medical Center Fargo, Fargo, North Dakota
  - 8400682 - Trinity Medical Group, Minot, North Dakota
  - 8400657 - Summa Health, Akron, Ohio
  - 8400793 - Aultman Hospital, Canton, Ohio
  - 8400858 - University of Cincinnati, Cincinnati, Ohio
  - 8401233 - Cincinnati V.A. Medical Center, Cincinnati, Ohio
  - 8400966 - MetroHealth System, Cleveland, Ohio
  - 8400565 - Miami Valley Hospital, Dayton, Ohio
  - 8400654 - North Ohio Research Ltd., Elyria, Ohio
  - 8400632 - North Ohio Heart Center, Sandusky, Ohio
  - 8400700 - Mercy Saint Vincent Medical Center, Toledo, Ohio
  - 8401164 - University of Toledo Medical Center, Toledo, Ohio
  - 8400639 - Genesis Health Care System, Zanesville, Ohio
  - 8400504 - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - 8400936 - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - 8400664 - Oklahoma Heart Institute, Tulsa, Oklahoma
  - 8401042 - Abington Medical Specialists, Abington, Pennsylvania
  - 8400595 - Lehigh Valley Hospital, Allentown, Pennsylvania
  - 8400608 - Holy Spirit Cardiology, Camp Hill, Pennsylvania
  - 8400872 - Chambersburg Hospital, Chambersburg, Pennsylvania
  - 8400577 - Doylestown Cardiology Associates, Doylestown, Pennsylvania
  - 8400324 - Milton Hershey Medical Center, Hershey, Pennsylvania
  - 8400344 - Lancaster General Hospital, Lancaster, Pennsylvania
  - 8400746 - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - 8400718 - V.A. Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - 8400570 - Advanced Cardiology Specialists, Scranton, Pennsylvania
  - 8401179 - Reading Hospital, West Reading, Pennsylvania
  - 8400794 - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - 8400811 - Rhode Island Hospital, Providence, Rhode Island
  - 8400591 - AnMed Health Medical Center, Anderson, South Carolina
  - 8401171 - Greenville Hospital System, Greenville, South Carolina
  - 8401055 - Upstate Cardiology, PA, Greenville, South Carolina
  - 8400496 - Advanced Cardiology Associates, Greenwood, South Carolina
  - 8400582 - Carolina Heart Specialists, Lancaster, South Carolina
  - 8400320 - Black Hills Cardiovascular Research, Rapid City, South Dakota
  - 8400854 - The Chattanooga Heart Institute, Chattanooga, Tennessee
  - 8400500 - Tennova Health Care - Turkey Creek Medical Center, Knoxville, Tennessee
  - 8400760 - V.A. Medical Center - Memphis, Memphis, Tennessee
  - 8400873 - Baptist Clinical Research Institute, Memphis, Tennessee
  - 8400801 - Centennial Medical Center, Nashville, Tennessee
  - 8400735 - Parkway Cardiology Associates, PC, Oak Ridge, Tennessee
  - 8400551 - Cardiovascular Research of Knoxville, Powell, Tennessee
  - 8400805 - PharmaTex Research, Amarillo, Texas
  - 8400482 - Amarillo Heart Clinical Research Institute, Amarillo, Texas
  - 8400485 - V.A. North Texas Health Care System, Dallas, Texas
  - 8400911 - Brooke Army Medical Center, Fort Sam Houston, Texas
  - 8401231 - Revival Research Institute, McKinney, Texas
  - 8400881 - North Texas Research Associates, McKinney, Texas
  - 8400921 - Mission Research Institute, LLC, New Braunfels, Texas
  - 8400704 - South Texas CV Consultants, San Antonio, Texas
  - 8400890 - Revival Research Institute, LLC, Sherman, Texas
  - 8401176 - Methodist Sugar Land Hospital, Sugar Land, Texas
  - 8400521 - CAET Research, Tyler, Texas
  - 8401128 - Hillcrest Family Health Center, Waco, Texas
  - 8400515 - Wichita Falls Heart Clinic, Wichita Falls, Texas
  - 8401064 - Inova Fairfax Hospital, Falls Church, Virginia
  - 8400502 - Stroobants Cardiovascular Center, Lynchburg, Virginia
  - 8400601 - McGuire Research Institute, Richmond, Virginia
  - 8400759 - Winchester Cardiology and Vascular Medicine, Winchester, Virginia
  - 8400628 - Multicare Health System, Puyallup, Washington
  - 8400863 - Swedish Medical Center - Providence Campus, Seattle, Washington
  - 8400503 - The Heart and Vascular Center / Holy Family Memorial, Manitowoc, Wisconsin
  - 8400358 - Aspirus Research Institute, Wausau, Wisconsin
- Argentina (32):
  - 0320069 - Hospital Italiano Regional del Sur, Bahía Blanca
  - 0320020 - Clinica Privada, Buenos Aires
  - 0320025 - Fundación Sanatorio Güemes, Ciudad Autonoma Buenos Aires
  - 0320041 - Clinica y Maternidad Suizo Argentina (CyMSA), Ciudad Autónoma Buenos Aires
  - 0320019 - Hospital Británico de Buenos Aires, Ciudad Autónoma Buenos Aires
  - 0320029 - Instituto Cardiovascular de Buenos Aires, Ciudad Autónoma Buenos Aires
  - 0320034 - Clinica Adventista Belgrano, Ciudad Autónoma Buenos Aires
  - 0320033 - Corporacion Medica de San Martin, Ciudad Autónoma Buenos Aires
  - 0320013 - Hospital Municipal de Coronel Suárez, Coronel Suárez
  - 0320040 - Instituto de Cardiología de Corrientes, Corrientes
  - 0320015 - Clinica Chutro S.R.L., Córdoba
  - 0320063 - Clinica Romagosa, Córdoba
  - 0320023 - Clínica Privada del Prado, Córdoba
  - 0320012 - Sanatorio Allende, Córdoba
  - 0320036 - Hospital Italiano, Córdoba
  - 0320026 - Clínica Colombo, Córdoba
  - 0320039 - Santatorio Parque S.A., Córdoba
  - 0320014 - Hospital Italiano La Plata, La Plata
  - 0320016 - Sanatorio Modelo Quilmes, Quilmes
  - 0320044 - Instituto Medico de la Fundacion de Estudios Clínicos, Rosario
  - 0320017 - Entidades Vinculadas al Sanatorio Parque, Rosario
  - 0320071 - Hospital Provincial del Centenario, Rosario
  - 0320070 - Hospital Papa Francisco, Salta
  - 0320073 - Instituto Medico De Alta Complejidad - IMAC, Salta
  - 0320022 - Hospital El Cruce, San Juan Bautista
  - 0320037 - Centro Privado de Cardiologia (CPC), San Miguel de Tucumán
  - 0320027 - Estudios Clínicos de los Arroyos, San Nicolás
  - 0320021 - Sanatorio Medico de Diagnostico y Tratamiento S.A., Santa Fe
  - 0320038 - Sanatorio Mayo Privado S.A., Santa Fe
  - 0320032 - Hospital Dr. Jose Maria Cullen, Santa Fe
  - 0320067 - Sanatorio Santa Rosa, Santa Rosa
  - 0320054 - Clínica Privada de Especialidades Médicas de Villa María, Villa María
- Australia (21):
  - 0360087 - Campbelltown Hospital, Campbelltown, New South Wales
  - 0360069 - Liverpool Hospital, Liverpool, New South Wales
  - 0360070 - Royal North Shore Hospital, St Leonards, New South Wales
  - 0360071 - Wollongong Hospital, Wollongong, New South Wales
  - 0360063 - Cairns Base Hospital, Cairns, Queensland
  - 0360062 - The Prince Charles Hospital, Chermside, Queensland
  - 0360061 - Royal Brisbane Hospital, Herston, Queensland
  - 0360060 - Gold Coast Hospital, Southport, Queensland
  - 0360057 - Royal Adelaide Hospital, Adelaide, South Australia
  - 0360032 - Flinders Medical Centre, Bedford Park, South Australia
  - 0360055 - Queen Elizabeth Hospital, Woodville South, South Australia
  - 0360084 - Royal Hobart Hospital, Hobart, Tazmania
  - 0360092 - Monash Medical Centre, Clayton, Victoria
  - 0360036 - The Northern Hospital, Epping, Victoria
  - 0360096 - Peninsula Health, Frankston, Victoria
  - 0360076 - Geelong Hospital, Geelong, Victoria
  - 0360081 - Peninsula Heart Centre, Langwarrin, Victoria
  - 0360073 - The Alfred Hospital, Melbourne, Victoria
  - 0360080 - Fiona Stanley Hospital, Murdoch, Western Australia
  - 0360059 - Royal Perth Hospital, Perth, Western Australia
  - 0360072 - John Hunter Hospital, New Lambton Heights
- Austria (5):
  - 0400035 - Landeskrankenhaus Feldkirch, Feldkirch
  - 0400020 - LKH-Universität Hospital Graz, Graz
  - 0400028 - Medizinische Universitaet Innsbruck - Universitaetsklinik für Innere Medizin, Innsbruck
  - 0400034 - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - 0400031 - Universitatsklinik fuer Innere Medizin II, Kardiol, Salzburg
- Belgium (22):
  - 0560024 - Onze-Lieve-Vrouwziekenhuis VZW (OLV), Aalst
  - 0560043 - Algemeen Stedelijk Ziekenhuis, Aalst
  - 0560027 - ZNA Middelheim, Antwerp
  - 0560028 - AZ Klina, Brasschaat
  - 0560020 - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - 0560015 - Clinique Saint Jean, Brussels
  - 0560023 - Centre Hospitalier Universitaire Brugmann, Brussels
  - 0560016 - Ziekenhuis Oost-Limburg, Genk
  - 0560037 - Universitair Ziekenhuis Gent, Ghent
  - 0560045 - AZ Sint-Lucas, Ghent
  - 0560038 - Jessa Ziekenhuis, Hasselt
  - 0560019 - Centre Hospitalier Régional de Huy, Huy
  - 0560026 - Universitair Ziekenhuis Brussel, Jette
  - 0560046 - AZ Groeninge - Campus Kennedylaan, Kortrijk
  - 0560022 - Centre Hospitalier Universitaire de Tivoli, La Louvière
  - 0560036 - Universitair Ziekenhuis Leuven, Leuven
  - 0560017 - CHR de la Citadelle, Liège
  - 0560053 - AZ Sint-Maarten, Mechelen
  - 0560044 - Heilig Hartziekenhuis Mol, Mol
  - 0560032 - AZ Delta, Roeselare
  - 0560018 - AZ Glorieux, Ronse
  - 0560040 - Campus Saint Elizabeth, Turnhout
- Brazil (41):
  - 0760069 - Hospital Universitario Evangelico de Curitiba, Curitiba, Paraná
  - 0760087 - MK BC Pesquisa Clinica, Balneário Camboriú
  - 0760056 - Hospital Felício Rocho, Belo Horizonte
  - 0760068 - Gutierrez Cardiologia Clinica e Intervencionista Ltda., Belo Horizonte
  - 0760085 - Hospital Universitário São José (HUSJ), Belo Horizonte
  - 0760021 - Fundacao Hospitalar Sao Francisco de Assis, Belo Horizonte
  - 0760059 - Hospital do Coração do Brasil, Brasília
  - 0760038 - Instituto de Cardiologia do Distrito Federal (ICDF), Brasília
  - 0760057 - Centro de Cardiologia Clinica e Pesquisa Dra. Juliana Souza, Brasília
  - 0760060 - Hospital Angelina Caron, Campina Grande do Sul
  - 0760077 - Instituto de Pesquisa Clinica de Campinas, Campinas
  - 0760035 - Loema - Instituto de Pesquisa Clinica, Campinas
  - 0760034 - Hospital e Maternidade Celso Pierro, Campinas
  - 0760061 - Hospital Universitario Maria Aparecida Pedrossian, Campo Grande
  - 0760036 - Hospital Geral Universitário de Cuiabá - HGU, Cuiabá
  - 0760011 - Hospital Cardiologico Costantini, Curitiba
  - 0760037 - Hospital de Messejana Dr. Carlos Alberto Gomes Studart, Fortaleza
  - 0760009 - Santa Casa de Misericordia de Marilia, Marília
  - 0760058 - Hospital São Vicente de Paulo, Passo Fundo
  - 0760040 - Santa Casa de Misericordia de Pelotas, Pelotas
  - 0760019 - Hospital São Lucas da PUCRS, Porto Alegre
  - 0760012 - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre
  - 0760015 - Hospital de Clínicas de Porto, Porto Alegre
  - 0760052 - Hospital Nossa Senhora da Conceicao (HNSC), Porto Alegre
  - 0760018 - Pronto Socorro Cardiológico de Pernambuco (PROCAPE), Recife
  - 0760062 - Hospital Agamenon Magalhães, Recife
  - 0760075 - Instituto D'Or de Pesquisa e Ensino, Rio de Janeiro
  - 0760025 - Hospital Santa Izabel, Salvador
  - 0760055 - Instituto Cardio Pulmonar da Bahia - Hospital, Salvador
  - 0760053 - Fundação Bahiana de Cardiologia, Salvador
  - 0760044 - Hospital da Bahia, Salvador
  - 0760041 - Hospital e Maternidade Dr. Christovao da Gama, Santo André
  - 0760027 - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - 0760047 - Instituto de Cardiologia de Santa Catarina (ICSC), São José
  - 0760016 - Faculdade de Medicina de Sao Jose do Rio Preto-SP - Hospital, São José do Rio Preto
  - 0760083 - Irmandade da Santa Casa de Misericordia de Sao Paulo, São Paulo
  - 0760031 - Instituto do Coração (InCor), São Paulo
  - 0760010 - Eurolatino Medical Research, Uberlândia
  - 0760039 - Hospital Evangelico de Vila Velha (HEVV), Vila Velha
  - 0760081 - Hospital Universitário Cassiano Antonio Moraes (HUCAM), Vitória
  - 0760028 - Santa Casa de Votuporanga, Votuporanga
- Bulgaria (21):
  - 1000023 - MHAT "Pulse AD", Blagoevgrad
  - 1000043 - Multiprofile Hospital for Active Treatment Blagoevgrad AD, Blagoevgrad
  - 1000074 - "UMHAT Deva Mariya" EOOD, Burgas
  - 1000072 - Multiprofile Hospital for Active Treatment - Dobrich AD, Dobrich
  - 1000029 - Multiprofile Hospital for Active Treatment AD Haskovo, Haskovo
  - 1000045 - MHAT City Clinic - Sv. Georgi EOOD, Lom
  - 1000036 - MHAT-Higia, Pazardzhik
  - 1000053 - Multiprofile Hospital For Active Treatment - Pazardzhik AD, Pazardzhik
  - 1000049 - SHATC Sv. Georgi - Pernik, Pernik
  - 1000071 - University Multiprofile Hospital for Active Treatment "Dr. G", Pleven
  - 1000057 - Specialized Hospital for Active Treatment in Cardiology EAD, Pleven
  - 1000058 - Multiprofile Hospital for Active Treatment Plovdiv AD, Plovdiv
  - 1000044 - Second Multiprofile Hospital for Active Treatment - Sofia EA, Sofia
  - 1000054 - Multiprofile Hospital for Active Treatment "National Cardiac Hospital", Sofia
  - 1000070 - University Multiprofile Hospital for Active Treatment Alexa, Sofia
  - 1000033 - University Multiprofile Hospital for Active Treatment, Sofia
  - 1000047 - University Hospital for Active Treatment & Emergency Medicine, Sofia
  - 1000035 - "MHAT "Sveta Anna"" - Sofia AD, Sofia
  - 1000038 - Acibadem City Clinic University Hospital, EOOD, Sofia
  - 1000028 - SHAT Cardiology Varna - EAD, Varna
  - 1000024 - Multiprofile District Hospital, Veliko Tarnovo
- Canada (33):
  - 1240063 - Heritage Medical Research Clinic, Calgary, Alberta
  - 1240032 - Royal Alexandra Hospital, Edmonton, Alberta
  - 1240058 - University of Alberta Hospital, Edmonton, Alberta
  - 1240074 - Vancouver General Hospital, Vancouver, British Colombia
  - 1240102 - Royal Inland Hospital, Kamloops, British Columbia
  - 1240101 - Kelowna General Hospital, Kelowna, British Columbia
  - 1240068 - Fraser Clinical Trials, Inc., New Westminster, British Columbia
  - 1240061 - SMH Cardiology Clinical Trials Inc., Surrey, British Columbia
  - 1240062 - Saint Boniface General Hospital, Winnipeg, Manitoba
  - 1240090 - New Brunswick Heart Centre Research Initiative, Saint John, New Brunswick
  - 1240060 - Health Sciences Centre, St. John's, Newfoundland and Labrador
  - 1240096 - William Osler Health System, Brampton, Ontario
  - 1240065 - Hamilton Health Sciences, Hamilton, Ontario
  - 1240091 - Kingston General Hospital, Kingston, Ontario
  - 1240069 - York PCI Group, Inc., Newmarket, Ontario
  - 1240093 - Halton Healthcare - Oakville Trafalgar Memorial Hospital, Oakville, Ontario
  - 1240077 - Ottawa Heart Institute, Ottawa, Ontario
  - 1240078 - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - 1240113 - Niagara Health System, St. Catherines Site, St. Catharines, Ontario
  - 1240097 - St. Michael's Hospital, Toronto, Ontario
  - 1240107 - Clinique de Cardiologie de Levis, Lévis, Quebec
  - 1240088 - Montreal Heart Institute, Montreal, Quebec
  - 1240092 - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - 1240106 - McGill University Health Centre (MUHC), Montreal, Quebec
  - 1240083 - CHU de Quebec-Universite-Laval, HDQ, Québec, Quebec
  - 1240099 - Centre Hospital Saint Georges de Beauce, Saint-Georges, Quebec
  - 1240081 - Saint Jerome Medical Research, Inc., Saint-Jérôme, Quebec
  - 1240087 - CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec
  - 1240059 - Centre Hospitalier Pierre-Le Gardeur, Terrebonne, Quebec
  - 1240066 - Centre Integre Universitaire de la Mauricie-et-du-Centre-du-Quebec, Trois-Rivières, Quebec
  - 1240095 - Royal University Hospital, Saskatoon, Saskatchewan
  - 1240071 - Institut universitaire de cardiologie et de pneumologie de Quebec, Québec
  - 1240079 - Toronto General Hospital, Toronto
- Chile (5):
  - 1520014 - Hospital Clinico Regional Dr. Guillermo Grant Benavente, Concepción
  - 1520017 - Hospital San Juan de Dios, Santiago
  - 1520026 - Hospital Las Higueras, Talcahuano
  - 1520004 - Hospital Dr. Hernan Henriquez Aravena, Temuco
  - 1520013 - Hospital de Victoria, Victoria
- Colombia (11):
  - 1700007 - Fundacion Cardiomet Eje Cafetero CEQUIN, Armenia
  - 1700008 - Clinica de la Costa, Barranquilla
  - 1700006 - Hospital Universitario San Ignacio, Bogotá
  - 1700011 - Fundación Valle del Lili, Cali
  - 1700010 - Centro Medico Imbanaco, Cali
  - 1700017 - Fundación Cardiovascular de Colombia, Floridablanca
  - 1700012 - Fundación Oftalmológica de Santander - Clinica FOSCAL, Floridablanca
  - 1700018 - Caja de Compensacion Familiar de Caldas, Manizales
  - 1700013 - Rodrigo Botero SAS, Medellín
  - 1700015 - Hospital Pablo Tobon Uribe, Medellín
  - 1700024 - Fundación Hospitalaria San Vicente de Paul, Medellín
- Croatia (6):
  - 1910010 - Županijska Bolnica Cakovec, Čakovec
  - 1910008 - Specijalna Bolnica za Medicinsku Rehabilitaciju Krapinske Toplice, Krapinske Toplice
  - 1910019 - Klinicki Bolnicki Centar Rijeka - Susak, Rijeka
  - 1910003 - Klinicki Bolnicki Centar Zagreb, Zagreb
  - 1910012 - Klinička Bolnica Sveti Duh, Zagreb
  - 1910013 - Klinički bolnički centar Sestre milosrdnice, Zagreb
- Czechia (13):
  - 2030048 - Fakultní Nemocnice Brno, Brno
  - 2030057 - Fakultní Nemocnice Hradec Králové, Hradec Králové
  - 2030031 - Nemocnice Jablonec nad Nisou, p.o., Jablonec nad Nisou
  - 2030073 - Karlovarska Krajska Nemocnice a.s., Karlovy Vary
  - 2030040 - Oblastní Nemocnice Kladno, a.s., Kladno
  - 2030061 - Oblastní nemocnice Náchod, a.s, Náchod
  - 2030041 - Nemocnice Pardubickeho kraje, a.s. - Pardubicka nemocnice, Pardubice
  - 2030020 - Fakultní nemocnice Královské Vinohrady, Prague
  - 2030038 - Vseobecna Fakultni Nemocnice, Ustav hematologie a krevni transfuze, Prague
  - 2030052 - Všeobecná fakultní nemocnice v Praze, Prague
  - 2030071 - Ústřední vojenská nemocnice - Vojenská fakultní nemocnice Praha, Prague
  - 2030050 - Nemocnice Slaný, Slaný
  - 2030059 - Uherskohradišťská nemocnice a.s., Uherské Hradiště
- Denmark (12):
  - 2080012 - Aalborg Universitetshospital, Aalborg
  - 2080022 - Amager Sygehus - Kardiologisk Klinik, Copenhagen
  - 2080009 - Sydvestjysk Sygehus - Esbjerg, Esbjerg
  - 2080021 - Amager and Hvidovre Hospital - Medical Department, Glostrup Municipality
  - 2080011 - Gentofte Hospital, Hellerup
  - 2080016 - Medicinsk Afdeling - Herning Sygehus, Herning
  - 2080008 - Hvidovre Hospital, Hvidovre
  - 2080015 - Koege Sygehus - University Hospital Sjaelland, Køge
  - 2080019 - Sjaellands Universitetshospital - Kardiologisk Afdeling, Roskilde
  - 2080018 - Regionshospitalet Silkeborg, Silkeborg
  - 2080014 - Svendborg Sygehus, Ward "Forskningsenheden Afd M Svendborg", Svendborg
  - 2080020 - Hjertesygdomme | Regionshospitalerne i Viborg og Skive, Viborg
- Estonia (3):
  - 2330006 - East-Tallinn Central Hospital, Tallinn
  - 2330005 - North Estonia Medical Centre Foundation, Tallinn
  - 2330004 - Tartu University Hospital, Tartu
- Finland (2):
  - 2460006 - Helsinki University Central Hospital (HUCH), Helsinki
  - 2460011 - Turku University Hospital (TYKS), Turku
- France (21):
  - 2500081 - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - 2500163 - CHU Caen, Caen
  - 2500162 - CHRU de Tours - Hopital Trousseau, Chambray-lès-Tours
  - 2500107 - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - 2500103 - CHU de Grenoble, Grenoble
  - 2500078 - Centre Hospitalier Louis Pasteur, Le Coudray
  - 2500117 - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - 2500112 - Centre Hospitalier Régional Universitaire de Lille (CHRU), Lille
  - 2500082 - Clinique du Pont de Chaume, Montauban
  - 2500091 - CHRU Montpellier - Arnaud de Villeneuve, Montpellier
  - 2500110 - CHU de Nantes, Nantes
  - 2500079 - CHU de Nice - Hôpital Pasteur, Nice
  - 2500105 - CHU de Nimes - Hopital Universitaire Caremeau, Nîmes
  - 2500090 - Hôpital Lariboisière, Paris
  - 2500046 - Hopital Pitie-Salpetriere, Paris
  - 2500101 - Hopital Paris Saint Joseph, Paris
  - 2500042 - CHU Hopitaux de Bordeaux - Hôpital Haut-Lévêque, Pessac
  - 2500165 - CHU de Poitiers, Poitiers
  - 2500120 - Centre Hospitalier Annecy Genevois, Pringy
  - 2500092 - Centre Hospitalier Régional Metz-Thionville, Thionville
  - 2500080 - CHU de Toulouse - Hopital Rangueil - Cardiologie, Toulouse
- Georgia (11):
  - 2680018 - TSMU - Alexandre Aladashvili University Clinic, Tbilisi
  - 2680002 - Helsicore - Israeli Georgian Medical Research Clinic, Tbilisi
  - 2680020 - Cardiological Clinic "Guli", Tbilisi
  - 2680004 - Clinical Cardology Institute Ltd., Tbilisi
  - 2680012 - Chapidze Emergency Cardiology Center, Tbilisi
  - 2680013 - Tbilisi Heart and Vascular Clinic LTD, Tbilisi
  - 2680015 - Chapidze Emergency Cardiology Center, Tbilisi
  - 2680026 - Georgian-Dutch Hospital MEDISON, Tbilisi
  - 2680010 - MediClub Georgia, Tbilisi
  - 2680027 - Tbilisi State Medical University (TSMU) - S. Khechinashvili, Tbilisi
  - 2680023 - LTD "Samgori Medi", Tbilisi
- Germany (27):
  - 2760133 - SLK - Klinikum am Plattenwald, Bad Friedrichshall
  - 2760143 - Vivantes Klinikum Am Urban, Berlin
  - 2760184 - Praxis Dr. Med. Nicole Toursarkissian, Berlin
  - 2760170 - Charite - UB - CVK - Medizinische Klinik, Berlin
  - 2760146 - Innere Medizin I, Marienhaus Klinikum Eifel Bitburg, Bitburg
  - 2760155 - Universitätsklinikum Bonn, Bonn
  - 2760141 - Klinikum Coburg GmbH, Coburg
  - 2760139 - Staedtisches Klinikum Dresden-Friedrichstadt - I. Medizinisc, Dresden
  - 2760243 - HELIOS Klinikum Erfurt, Erfurt
  - 2760164 - Elisabeth-Krankenhaus Essen GmbH Klinik für Kardiologie und Angiologie, Essen
  - 2760193 - CardioVaskulares Centrum Frankfurt, Frankfurt am Main
  - 2760168 - Klinikum Frankfurt Höchst GmbH, Frankfurt am Main
  - 2760119 - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - 2760219 - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - 2760190 - Asklepios Kliniken Hamburg GmbH, Hamburg
  - 2760140 - Cardiologicum Hamburg - Studienzentrum, Hamburg
  - 2760188 - Asklepios Klinik Barmbek, Hamburg
  - 2760149 - Asklepios Klinik Altona, Hamburg
  - 2760135 - University Hospital Jena, Jena
  - 2760132 - Ambulantes Herzzentrum Kassel, Kassel
  - 2760181 - Asklepios Klinik Langen, Langen
  - 2760111 - Klinikum der Stadt Ludwigshafen gGmbH, Ludwigshafen
  - 2760130 - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - 2760186 - Katholisches Klinikum Mainz - Klinik fuer Innere Medizin I, Mainz
  - 7240030 - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - 2760147 - GPR Klinikum Rüsselsheim II - Medizinische Klinik Innere Medizin, Rüsselsheim am Main
  - 2760176 - Evangelisches Krankenhaus Witten, Witten
- Greece (11):
  - 3000027 - GENERAL HOSPITAL Korgialenio - Benakio HRC, Athens
  - 3000022 - University of Athens - Hippokration General Hospital, Athens
  - 3000023 - National and Kapodistrian University of Athens (NKUA) - Scho, Athens
  - 3000026 - University General Hospital Attikon, Chaïdári
  - 3000016 - General Hospital of Thessaloniki "G. Papanikolaou", Chortiatis
  - 3000008 - University of Ioannina School of Medicine - Michaelidion Cardiac Center, Ioannina
  - 3000010 - University Hospital of Ioannina, Ioannina
  - 3000029 - University of Thessaly- General University Hospital of Laris, Larissa
  - 3000025 - University General Hospital of Patras, Pátrai
  - 3000007 - General Hospital of Nikea "Agios Panteleimon", Piraeus
  - 3000013 - University General Hospital of Thessaloniki AHEPA, Thessaloniki
- Hong Kong (3):
  - 3440004 - Queen Elizabeth Hospital (QEH), Kowloon
  - 3440005 - Princess Margaret Hospital, Kwai Chung
  - 3440006 - Prince of Wales Hospital, Shatin
- Hungary (17):
  - 3480016 - Budai Irgalmasrendi Kórház, Budapest
  - 3480024 - Bajcsy-Zsilinszky Hospital, Budapest
  - 3480033 - Semmelweis University, Faculty of Medicine, Budapest
  - 3480028 - Magyar Honvédség Egészségügyi Központ, Budapest
  - 3480040 - Jahn Ferenc Dél-pesti Kórház és Rendelőintézet, Budapest
  - 3480019 - Debreceni Egyetem Klinikai Központ, Debrecen
  - 3480025 - Dombovari Szent Lukacs Egeszsegugyi Kft, Dombóvár
  - 3480023 - Petz Aladar County Teaching Hospital, Győr
  - 3480029 - Békés Megyei Pándy Kálmán Kórház, Gyula
  - 3480045 - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
  - 3480036 - Bács-Kiskun Megyei Kórház, Kecskemét
  - 3480015 - Jósa András Oktatókórház, Nyíregyháza
  - 3480022 - University of Szeged - Second Department of Medicine & Cardiology Centre, Szeged
  - 3480035 - Tolna Megyei Balassa Janos Korhaz, Szekszárd
  - 3480020 - Fejér Megyei Szent György Egyetemi Oktató Kórház, Székesfehérvár
  - 3480018 - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház-Rendelőintéz, Szolnok
  - 3480026 - Zala Megyei Szent Rafael Kórház, Zalaegerszeg
- Israel (21):
  - 3760021 - Emek Medical Center, Afula
  - 3760041 - Emek Medical Center, Afula
  - 3760028 - Barzilai Medical Center, Ashkelon
  - 3760024 - Soroka Medical Center, Beersheba
  - 3760034 - Assaf Harofeh Medical Center - Cardiology Division, Be’er Ya‘aqov
  - 3760032 - Hillel Yaffe Medical Center, Hadera
  - 3760022 - Bnai Zion Medical Center, Haifa
  - 3760014 - Rambam Medical Center, Haifa
  - 3760012 - Hadassah Ein Karem Hospital, Jerusalem
  - 3760023 - Shaare Zedek Medical Center, Jerusalem
  - 3760029 - Hadassah Medical Center-Mount Scopus, Jerusalem
  - 3760037 - Tel Aviv University Sackler School of Medicine - Meir Medica, Kfar Saba
  - 3760020 - Galilee Medical Center, Nahariya
  - 3760026 - The Baruch Padeh Medical Center, Nazareth
  - 3760035 - The Baruch Padeh Medical Center, Nazareth
  - 3760025 - Rabin Medical Center - Hasharon Hospital, Petah Tikva
  - 3760018 - Leviev Heart Center, Chaim Sheba Medical Center, Ramat Gan
  - 3760027 - Kaplan Medical Center, Rehovot
  - 3760019 - Ziv MC, Safed
  - 3760036 - Assuta Medical Center, Tel Aviv
  - 3760038 - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (17):
  - 3800062 - ASST Papa Giovanni XXIII, Bergamo
  - 3800075 - ASST degli Spedali Civili di Brescia, Brescia
  - 3800170 - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - 3800085 - Azienda Socio-Sanitaria Territoriale della Valle Olona, Busto Arsizio
  - 3800079 - Azienda Ospedaliera di Caserta "Sant'Anna e San Sebastiano", Caserta
  - 3800107 - Università degli Studi "Magna Graecia" di Catanzaro, Catanzaro
  - 3800129 - Azienda Ospedaliero-Universitaria Careggi, Florence
  - 3800141 - IRCCS MultiMedica, Milan
  - 3800088 - Centro Cardiologico Monzino, Milan
  - 3800087 - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - 3800123 - AORN - Ospedali dei Colli Ospedale V. Monaldi, Napoli
  - 3800090 - Gruppo Ospedaliero San Donato - Policlinico San Marco, Osio Sotto
  - 3800082 - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - 3800110 - Fondazione IRCCS Policlinico San Matteo, Pavia
  - 3800080 - ASL Roma 2, Roma
  - 3800106 - Università degli Studi di Roma "La Sapienza", Roma
  - 3800056 - Istituto Clinico Humanitas, Rozzano
- Japan (38):
  - 3920154 - Kurashiki Central Hospital, Kurashiki-shi, Okayama-ken
  - 3920130 - Eiyukai Ayase Heart Hospital, Adachi-Ku
  - 3920106 - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki-Shi
  - 3920095 - Showa University Fujigaoka Hospital, Aoba-Ku
  - 3920156 - Asahi General Hospital, Asahi-Shi
  - 3920122 - Sakakibara Heart Institute, Fuchu-Shi
  - 3920105 - Fukuoka University Hospital, Fukuoka
  - 3920101 - Teikyo University Hospital, Itabashi-Ku
  - 3920116 - Nihon University Itabashi Hospital, Itabashi-Ku
  - 3920094 - Juntendo University Shizuoka Hospital, Izunokuni-Shi
  - 3920111 - Ishikawa Prefectural Central Hospital, Kanazawa
  - 3920108 - Fukuoka Tokushukai Hospital, Kasuga-Shi
  - 3920134 - Kimitsu Chuo Hospital, Kisarazu-Shi
  - 3920092 - Chikamori Hospital, Kochi
  - 3920109 - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - 3920113 - Kumamoto University Hospital, Kumamoto
  - 3920100 - Saiseikai Kumamoto Hospital, Kumamoto
  - 3920110 - Kurume University Hospital, Kurume-Shi
  - 3920136 - Shin Koga Hospital, Kurume-Shi
  - 3920103 - Kusatsu General Hospital, Kusatsu-Shi
  - 3920115 - Matsusaka Chuo General Hospital, Matsusaka-Shi
  - 3920119 - Ehime Prefectural Central Hospital, Matsuyama
  - 3920114 - Toho University Ohashi Medical Center, Meguro-ku
  - 3920093 - Miyazaki Medical Association Hospital, Miyazaki
  - 3920107 - Teine Keijinkai Hospital, Sapporo
  - 3920118 - Sapporo Medical University Hospital, Sapporo
  - 3920121 - Hokkaido Cardiovascular Hospital, Sapporo
  - 3920149 - Tohoku University Hospital, Sendai
  - 3920117 - Sendai Open Hospital, Sendai
  - 3920132 - Tosei General Hospital, Seto-Shi
  - 3920123 - Tokyo Women's Medical University Hospital, Shinjuku-Ku
  - 3920104 - Shizuoka City Shizuoka Hospital, Shizuoka
  - 3920120 - National Cerebral and Cardiovascular Center, Suita-Shi
  - 3920126 - Kagawa Prefectural Hospital, Takamatsu
  - 3920102 - Oji General Hospital, Tomakomai-Shi
  - 3920128 - Tokyo Bay Urayasu Ichikawa Medical Center, Urayasu-Shi
  - 3920099 - Yokohama City University Medical Center, Yokohama
  - 3920133 - Kanagawa Cardiovascular and Respiratory Center, Yokohama
- Latvia (5):
  - 4280004 - Daugavpils Regional Hospital, Daugavpils
  - 4280007 - Liepajas Regionala Slimnica, Liepāja
  - 4280008 - Pauls Stradins Clinical University Hospital, Riga
  - 4280005 - SIA Rigas Austrumu Kliniska Universitates Slimnica - Gaileze, Riga
  - 4280003 - Vidzemes slimnīca, Valmiera
- Lithuania (5):
  - 4400004 - Hospital of Lithuanian University of Health Sciences - Kauno Klinikos, Kaunas
  - 4400007 - Klaipėda Seamen's Hospital, Klaipėda
  - 4400006 - Public Institution Republican Panevezys Hospital, Panevezys
  - 4400008 - Republican Šiauliai Hospital, Šiauliai
  - 4400005 - Vilnius University Hospital Santaros Klinikos, Vilnius
- Malaysia (9):
  - 4580004 - Queen Elizabeth Hospital II, Kota Kinabalu, Sabah
  - 4580015 - Hospital Universiti Sains Malaysia, Kota Bharu
  - 4580007 - Institut Jantung Negara, Kuala Lumpur
  - 4580008 - Universiti Kebangsaan Malaysia Medical Centre, Kuala Lumpur
  - 4580016 - University Malaya Medical Centre, Kuala Lumpur
  - 4580003 - Hospital Tengku Ampuan Afzan, Kuantan
  - 4580002 - Hospital Umum Sarawak (HUS) - The Cardiac Centre, Kuching
  - 4580019 - Hospital Pulau Pinang, Pulau Pinang
  - 4580005 - Universiti Teknologi MARA (UiTM), Sungai Buloh
- Mexico (20):
  - 4840008 - Hospital Civil de Guadalajara - Nuevo Hospital Civil de Guadalajara, Guadalajara, Jalisco
  - 4840014 - Investigacion Biomedica para el Desarrollo de Farmacos S.A d, Aguascalientes
  - 4840004 - Hospital Cardiológica Aguascal, Aguascalientes
  - 4840077 - Unidad de Investigacion en Salud (UIS), Chihuahua City
  - 4840046 - Unidad de Investigacion, Chihuahua City
  - 4840006 - Centro para el Desarrollo de la Medicina y de Asistencia Méd, Culiacán
  - 4840033 - Virgen Cardiovascular Research S.C., Guadalajara
  - 4840020 - Centro de Estudios de Alta Especialidad de Sinaloa, S.C., Mazatlán
  - 4840034 - Hospital de Jesus, Mexico City
  - 4840016 - Instituto Nacional de Cardiologia Ignacio Chavez, México
  - 4840045 - OCA Hospital - Monterrey International Research Center, Monterrey
  - 4840036 - Cardiolink Clin Trials, SC., Monterrey
  - 4840021 - Universidad Autonoma de Nuevo Leon - Hospital Universitario, Monterrey
  - 4840007 - Unidad de Prevención y Atención Cardiometabólica (UPAC), Morelia
  - 4840074 - Unidad de Investigación y Salud de Puebla S.C., Puebla City
  - 4840003 - Centro de Estudios Clínicos de Querétaro, SC, Querétaro
  - 4840022 - Centro de Atencion e Investigacion Cardiovascular del Potosi, San Luis Potosí City
  - 4840025 - Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City
  - 4840076 - CIMAB S.A. de C.V., Torreón
  - 4840018 - Centro de Alta Especialidad Dr. Rafael Lucio, Xalapa
- Netherlands (29):
  - 5280054 - Noordwest Ziekenhuisgroep - Alkmaar, Alkmaar
  - 5280031 - Meander Medisch Centrum - Locatie Amersfoort, Amersfoort
  - 5280057 - Bovenij ziekenhuis, Amsterdam
  - 5280039 - OLVG Location West, Amsterdam
  - 5280061 - Amsterdam UMC - VUMC, Amsterdam
  - 5280016 - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - 5280048 - Amphia Zienkenhuis - Locatie Molengracht Breda, Breda
  - 5280047 - Deventer Hospital, Deventer
  - 5280013 - Ziekenhuis Gelderse Vallei, Ede
  - 5280040 - Maxima Medisch Centrum, Eindhoven
  - 5280049 - Medisch Spectrum Twente, Enschede
  - 5280038 - Admiraal de Ruijter Ziekenhuis - Locatie Goes, Goes
  - 5280056 - Groene Hart Ziekenhuis - Gouda, Gouda
  - 5280034 - Spaarne Gasthuis, Haarlem
  - 5280052 - Ziekenhuis St Jansdal, Harderwijk
  - 5280063 - Zuyderland Medisch Centrum, Heerlen, Heerlen
  - 5280037 - Dijklander Ziekenhuis - Hoorn, Hoorn
  - 5280045 - Medisch Centrum Leeuwarden, Leeuwarden
  - 5280064 - Alrijne Ziekenhuis Leiden, Leiden
  - 5280043 - Radboud UMC, Nijmegen
  - 5280036 - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - 5280062 - Sint Franciscus Gasthuis, Rotterdam
  - 5280018 - Maasstad Ziekenhuis, Rotterdam
  - 5280035 - D & A Research, Sneek
  - 5280060 - Ziekenhuis Rivierenland - Cardiologie, Tiel
  - 5280042 - Elisabeth TweeSteden Ziekenhuis Vestiging Tilburg, Tilburg
  - 5280058 - Universitair Medisch Centrum Utrecht, Utrecht
  - 5280020 - VieCuri, Venlo
  - 5280046 - Gelre Ziekenhuizen - Zutphen, Zutphen
- New Zealand (8):
  - 5540010 - North Shore Hospital, Takapuna, Auckland
  - 5540011 - Wellington Hospital, Newtown, Wellington Region
  - 5540017 - Auckland City Hospital, Auckland
  - 5540004 - Middlemore Hospital, Auckland
  - 5540008 - Christchurch Hospital, Christchurch
  - 5540009 - Dunedin Hospital, Dunedin
  - 5540005 - Waikato Hospital, Hamilton
  - 5540007 - Taranaki Base Hospital, New Plymouth
- Norway (4):
  - 5780003 - Akershus Universitetssykehus HF, Lørenskog
  - 5780011 - Diakonhjemmet Sykehus, Oslo
  - 5780010 - Sykehuset Telemark HF - Skien, Skien
  - 5780006 - Helse Stavanger HF, Stavanger
- Peru (3):
  - 6040031 - Clínica Internacional - Sede San Borja, Lima
  - 6040056 - Instituto Nacional Cardiovascular - INCOR, Lima
  - 6040017 - Clinica El Golf, Lima
- Poland (24):
  - 6160082 - II Oddział Kardiologiczny PAKS, Bielsko-Biala
  - 6160063 - Klinika Kardiologii i Kardiochirurgii 10 WSK, Bydgoszcz
  - 6160081 - McSn, Chrzanów
  - 6160065 - III Oddział Kardiologii Inwazyjnej, Angiologii i Elektrokard, Dąbrowa Górnicza
  - 6160054 - SPS Szpital Zachodni, Grodzisk Mazowiecki
  - 6160066 - IV Oddział Kardiologii Inwazyjnej, Elektrostymulacji i Angio, Kędzierzyn-Koźle
  - 6160078 - Nowy Szpital Uniwersytecki w Krakowie-Prokocimiu, Krakow
  - 6160051 - Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow
  - 6160095 - Centrum Kardiologii Inwazyjnej i Angiologii w Krośnie, Krosno
  - 6160096 - 1 Wojskowy Szpital Kliniczny z Poliklinika SPZOZ w Lublinie, Lublin
  - 6160062 - Wielospecjalistyczny Szpital Samodzielny Publiczny Zakład Op, Nowa Sól
  - 6160064 - Medicome sp.zoo, Oświęcim
  - 6160100 - Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii, Pińczów
  - 6160077 - Samodzielny Publiczny Zakład Opieki Zdrowotnej w Puławach, Puławy
  - 6160088 - Ikardia, Puławy
  - 6160080 - Regional Public Specialty Hospital "Latawiec", Swidnica
  - 6160067 - Szpital Polski - Sztum, Sztum
  - 6160061 - Wojewódzki Szpital Zespolony im. Ludwika Rydygiera w Toruniu, Torun
  - 6160073 - American Heart of Poland, Tychy
  - 6160052 - Szpital Wolski, Warsaw
  - 6160075 - Szpital Bielanski, Warsaw
  - 6160086 - Dept. of Interventional cardiology and Angiology, Institute, Warsaw
  - 6160093 - Specjalistyczny Szpital im. dr Alfreda Sokolowskiego, Wałbrzych
  - 6160083 - Wojewódzki Szpital Specjalistyczny im. Marii Skłodowskiej-Curie, Zgierz
- Portugal (11):
  - 6200011 - Hospital Garcia de Orta, EPE, Almada
  - 6200026 - Centro Hospitalar do Baixo Vouga, Aveiro
  - 6200015 - Hospital de Braga, Braga
  - 6200018 - Centro Hospitalar e Universitário de Coimbra, EPE - Hospitai, Coimbra
  - 6200022 - Centro Hospitalar e Universitário de Coimbra, EPE - Hospital, Coimbra
  - 6200012 - Centro Hospitalar e Universitário do Algarve, EPE - Hospital, Faro
  - 6200021 - Centro Hospitalar do Alto Ave, EPE, Guimarães
  - 6200009 - Hospital de Santo Andre, Leiria
  - 6200014 - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital Santa, Oeiras
  - 6200025 - Unidade Local de Saude de Matosinhos - Hospital Pedro Hispan, Senhora da Hora
  - 6200017 - Centro Hospitalar de Trás-os-Montes e Alto Douro, EPE - Hospital, Vila Real
- Romania (20):
  - 6420052 - Spitalul Judeţean de Urgenţă "Dr. Constantin Opriş" Baia Mar, Baia Mare
  - 6420053 - Spitalul Clinic Judetean de Urgenta Brasov, Brasov
  - 6420046 - Spitalului Universitar de Urgenţă Militar Central "Dr. Carol Davila", Bucharest
  - 6420090 - Spitalul Clinic de Urgenţă "Bagdasar-Arseni", Bucharest
  - 6420043 - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - 6420050 - Spitalul Universitar de Urgent, Bucharest
  - 6420051 - Institutul Inimii "Niculae Stancioiu", Cluj-Napoca
  - 6420088 - Institutul Inimii "Niculae Stancioiu", Cluj-Napoca
  - 6420060 - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca
  - 6420080 - Spitalul Clinic de Recuperare Cluj-Napoca, Cluj-Napoca
  - 6420044 - Spitalul Clinic Judetean de Ur, Craiova
  - 6420057 - Institutul de Boli Cardiovasculare "Prof. Dr. George I. M. Georgescu, Iași
  - 6420045 - Spitalul Clinic Judeţean de Urgenţă Oradea, Oradea
  - 6420048 - Spitalul Judetean de Urgenta Pitesti-Arges, Piteşti
  - 6420079 - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
  - 6420047 - Spitalul de Urgenta "Sf. Ioan Cel Nou" Suceava, Suceava
  - 6420059 - Institutul de Urgenta pentru Boli Cardiovasculare si Transplant, Târgu Mureş
  - 6420049 - Spitalul Clinic Judetean de Urgenta Tîrgu - Mures, Târgu Mureş
  - 6420071 - Institutului de Boli Cardiovasculare Timişoara, Timișoara
  - 6420083 - Institutului de Boli Cardiovasculare Timişoara, Timișoara
- Russia (32):
  - 6430075 - First City Clinical Hospital named after E. E. Volosevich, Arkhangelsk
  - 6430069 - Regional Clinical Hospital, Barnaul
  - 6430060 - Regional State Budgetary Institution of Public Health, Barnaul
  - 6430068 - Regional Budgetary Healthcare Institution "Cardiology Dispensary", Ivanovo
  - 6430116 - City hospital # 2 "Sosnovaya roscha", Kaluga
  - 6430079 - Scientific-Research Institute of Complex Problems of Cardio, Kemerovo
  - 6430048 - City Clinical Hospital No. 6 named after Karpovicha, Krasnoyarsk
  - 6430050 - Kursk City Emergency Care Hospital, Kursk
  - 6430063 - Lyubertsy Regional Hospital No. 2, Lyubertsy
  - 6430105 - City Clinical Hospital No. 51, Moscow
  - 6430091 - City clinical hospital #15 n.a. O.M. Filatov, Moskva
  - 6430080 - City Clinical Hospital No. 5, Nizhny Novgorod
  - 6430110 - SBHI of Novosibirsk Region "City Clinical Hospital of Emergency Care #2", Novosibirsk
  - 6430058 - State Budget Healthcare Institution of Novosibirsk Region "C, Novosibirsk
  - 6430047 - Novosibirsk Regional Clinical Hospital, Novosibirsk
  - 6430045 - Penza Regional Clinical Hospital n.a. N.N.Burdenko, Penza
  - 6430054 - City Clinical Hospital No. 4, Perm
  - 6430064 - City Hospital for Emergency Care of Rostov-on-Don, Rostov-on-Don
  - 6430070 - Saint-Petersburg I.I. Dzhanelidze Research Institute of Emergency Medicine, Saint Petersburg
  - 6430074 - St. Petersburg State Institution of Healthcare, Saint Petersburg
  - 6430107 - Clinical Hospital of the Russian Academy of Science, Saint Petersburg
  - 6430081 - Saint Petersburg State Medical Academy, Saint Petersburg
  - 6430115 - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - 6430049 - Pokrovskaya Municipal Hospital, Saint Petersburg
  - 6430072 - Samara Regional Cardiology Dispensary, Samara
  - 6430067 - Saratov State Medical University named after V.I. Razumovsky, Saratov
  - 6430042 - Research Institute of Cardiology, Tomsk
  - 6430043 - Tula Regional Clinical Hospital, Tula
  - 6430053 - Tyumen Cardiology Center, Tyumen
  - 6430111 - Clinical Hospital No. 8, Yaroslavl
  - 6430092 - Yaroslavl Regional Clinical Hospital, Yaroslavl
  - 6430108 - Novaya Bolnitsa, Yekaterinburg
- Serbia (16):
  - 6880014 - Klinički Centar Srbije, Belgrade, Savski Venac
  - 6880008 - Clinical Center of Serbia -- Division of Cardiology, Belgrade
  - 6880009 - Department of Cardiology, Clinical Center of Serbia and Belgrade, Belgrade
  - 6880019 - KBC "Dr Dragiša Mišović-Dedinje", Belgrade
  - 6880023 - Kliničko Bolnički Centar Zvezdara, Belgrade
  - 6880012 - Institute of Cardiovascular Diseases of Vojvodina, Kamenitz
  - 6880010 - Klinički Centar Kragujevac, Kragujevac
  - 6880015 - General Hospital Leskovac, Leskovac
  - 6880016 - Klinički Centar Niš, Niš
  - 6880026 - Opšta Bolnica Pančevo, Pančevo
  - 6880018 - Klinički Centar Srbije, Savski Venac
  - 6880013 - General Hospital Sremska Mitrovica, Sremska Mitrovica
  - 6880027 - General Hospital Subotica, Subotica
  - 6880020 - Zdravstveni Centar Užice, Užice
  - 6880025 - General Hospital Valjevo, Valjevo
  - 6880024 - Opsta Bolnica "Dorde Joanovic" Zrenjanin, Zrenjanin
- Singapore (2):
  - 7020005 - National University Hospital (S) Pte Ltd, Singapore
  - 7020006 - National Heart Center Singapore, Singapore
- Slovakia (5):
  - 7030006 - Univerzitna Nemocnica Bratislava - Nemocnica Staré Mesto, Bratislava
  - 7030014 - Univerzitna Nemocnica Bratislava - Nemocnica sv. Cyrila a Me, Bratislava
  - 7030013 - Nemocnica Malacky, Malacky
  - 7030003 - Kardiocentrum Nitra s.r.o., Nitra
  - 7030002 - Svet zdravia, a.s. - Všeobecná nemocnica Rimavská Sobota, Rimavská Sobota
- South Africa (9):
  - 7100006 - Mediclinic Vergelegen, Somerset West, Cape Town
  - 7100022 - Mediclinic Vergelegen, Somerset West, Cape Town
  - 7100007 - Netcare Unitas Hospital, Lyttelton, Centurion
  - 7100012 - Netcare Unitas Hospital, Lyttelton, Centurion
  - 7100023 - Tread Research, Cape Town
  - 7100019 - Groote Schuur Hospital, Cape Town
  - 7100017 - Netcare Union Hospital, Johannesburg
  - 7100020 - Netcare Sunninghill Hospital, Sunninghill
  - 7100010 - Clinical Projects Research SA (Pty) Ltd., Worcester
- South Korea (14):
  - 4100013 - Kyung Hee University Medical Center, Hoegi-dong, Dongdaemun-gu
  - 4100020 - Kyung Hee University Hospital at Gangdong, Seoul, Gangdong-gu
  - 4100014 - Yonsei University, Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - 4100024 - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - 4100015 - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - 4100019 - Kangbuk Samsung Hospital, Seoul, Jongro-gu
  - 4100025 - Korea University Anam Hospital, Seoul, Seongbuk-gu
  - 4100021 - Chungbuk National University Hospital, Cheongju-si
  - 4100016 - Veterans Health Service Medical Center, Gangdong
  - 4100017 - Chungnam National University Hospital, Junggu
  - 4100008 - Seoul National University Hospital, Seoul
  - 4100018 - Asan Medical Center, Seoul
  - 4100010 - The Catholic University of Korea, St. Vincent's Hospital, Suwon
  - 4100022 - Hallym University Sacred Heart Hospital, Yeongdeungpo-dong
- Spain (16):
  - 7240035 - Complexo Hospitalario Universitario A Coruña, A Coruña
  - 7240043 - Hospital Universitario Fundación Alcorcón, Alcorcón
  - 7240064 - Hospital General Universitario de Alicante, Alicante
  - 7240062 - Hospital del Mar, Barcelona
  - 7240050 - Hospital de la Santa Creu i Sant Pau, Barcelona
  - 7240063 - Hospital Universitario Vall d'Hebron, Barcelona
  - 7240033 - Hospital Clínic de Barcelona, Barcelona
  - 7240076 - Hospital Juan Ramón Jiménez, Huelva
  - 7240053 - Hospital Universitari de Bellvitge (IDIBELL), L'Hospitalet de Llobregat
  - 7240077 - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - 7240045 - Hospital Universitario Ramón y Cajal, Madrid
  - 7240070 - Hospital Universitario Virgen Arrixaca, Murcia
  - 7240068 - Hospital Universitario Marqués de Valdecilla, Santander
  - 7240032 - Hospital Universitari Joan XXIII de Tarragona, Tarragona
  - 7240034 - Hospital Clinico Universitario de Valencia, Valencia
  - 7240100 - Hospital Álvaro Cunqueiro, Vigo
- Sweden (4):
  - 7520023 - Örebro University Hospital, Örebro
  - 7520024 - Ostersunds Sjukhus, Östersund
  - 7520011 - Karolinska Universitetssjukhuset - Huddinge, Stockholm
  - 7520015 - Västmanlands Sjukhus Västerås, Västerås
- Switzerland (3):
  - 7560025 - University Hospital, Basel
  - 7560014 - Cardiocentro Ticino, Lugano
  - 7560019 - Stadtspital Triemli, Zurich
- Taiwan (9):
  - 1580012 - Cheng Hsin General Hospital, Taipei, Beitou
  - 1580001 - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - 1580002 - Kaohsiung Veterans General Hospital, Kaohsiung City
  - 1580006 - E-Da Hospital, Kaohsiung City
  - 1580008 - Mackay Memorial Hospital - Tamsui Branch, New Taipei City
  - 1580010 - China Medical University Hospital, Taichung
  - 1580007 - Chi Mei Medical Center, Tainan
  - 1580004 - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - 1580009 - National Taiwan University Hospital, Zhongzheng
- Thailand (8):
  - 7640012 - Ramathibodi Hospital, Bangkok
  - 7640021 - Chiang Mai University, Chiang Mai
  - 7640017 - Khon Kaen University (KKU), Khon Kaen
  - 7640018 - Maharat Nakhon Ratchasima Hospital, Nakhon Ratchasima
  - 7640010 - King Chulalongkorn Memorial Hospital, Pathum Wan
  - 7640014 - Police General Hospital, Pathum Wan
  - 7640020 - Buddhachinaraj Hospital Phitsanuloke, Phitsanulok
  - 7640009 - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (14):
  - 7920024 - Afyon Kocatepe University Medical Faculty Dept. Of Cardiology, Afyonkarahisar
  - 7920030 - T. C. Saglık Bakanlıgı - Bagcılar Egitim ve Arastırma Hastan, Bağcılar
  - 7920018 - Cukurova University School Of Medicine Balcali Hospital, Balcalı
  - 7920023 - Ege Üniversitesi Tıp Fakültesi, Bornova
  - 7920016 - Ankara Sehir Hastanesi Bilkent, Çankaya
  - 7920021 - Istanbul Universitesi Istanbul Tip Fakultesi, Çapa
  - 7920017 - Eskişehir Osmangazi Üniversitesi Tıp Fakültesi, Eskişehir
  - 7920012 - Istanbul Universitesi Cerrahpasa Tip Fakultesi Hastanesi, Fatih
  - 7920022 - Marmara Universitesi Tip Fakultesi, Istanbul
  - 7920032 - Kocaeli Universitesi Tip Fakultesi - Kardiyoloji Anabilim Dalı Başkanı, Kocaeli
  - 7920015 - T.C. Saglik Bakanligi - Kartal Kosuyolu Yuksek Ihtisas Egitim, Maltepe
  - 7920014 - Mersin Üniversitesi Tip Fakültesi, Mersin
  - 7920026 - Ondokuz Mayis Üniversitesi - Kardiyoloji Anabilim Dalı, Samsun
  - 7920025 - Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi - Kardiyo, Yıldırım
- Ukraine (23):
  - 8040019 - Cherkasy Regional Cardiological Center, Cherkasy
  - 8040010 - Dnipropetrovsk Medical Academy, Dnipropetrovsk Joint Emergen, Dnipro
  - 8040037 - The Ivano-Frankivsk National Medical Univeristy, Ivano-Frankivsk
  - 8040032 - Ivano-Frankivskyy oblasnyy klinichnyy kardiologichnyy dyspan, Ivano-Frankivsk
  - 8040048 - Communal Institution of Healthcare "Kharkiv Municipal Clinic, Kharkiv
  - 8040017 - National Institute of Therapy named after L.T. Malaya NAMS o, Kharkiv
  - 8040050 - Regional Clinical Hospital - Emergency Medical Care, Kharkiv
  - 8040012 - Kharkiv City Clinical Hospital #8, Kharkiv
  - 8040013 - Khmelnytskyi Regional Hospital, Khmelnytskyi
  - 8040047 - Oleksandrivska Clinical Hospital, Kyiv
  - 8040008 - Kyiv City Clinical Hospital No. 1, Kyiv
  - 8040021 - Heart Institute of the Ministry of Health of Ukraine, Kyiv
  - 8040009 - Kiev City Clinical Hospital No. 5, Kyiv
  - 8040025 - National Scientific Center, Kyiv
  - 8040049 - Lutsk City Clinical Hospital, Lutsk
  - 8040016 - Lviv National Medical University named by Danylo Halitskyy, Lviv
  - 8040035 - Lviv Regional State Clinical-and-Diagnostic Cardiology Cente, Lviv
  - 8040038 - City Hospital 4, Mykolaiv
  - 8040014 - Odessa Regional Hospital, Odesa
  - 8040015 - Ternopil University Hospital, Ternopil
  - 8040020 - Uzhgorod National University, Uzhhorod
  - 8040036 - Regional Medical Center for Cardiovascular Diseases, Zaporizhzhia
  - 8040023 - Zhitomir Regional Clinical Hospital, Zhytomyr
- United Kingdom (15):
  - 8260102 - Queen Elizabeth Hospital Birmingham, Birmingham
  - 8260057 - Mid Essex Hospital Services NHS Trust - Broomfield Hospital, Chelmsford
  - 8260071 - Ashford and St Peter's Hospitals NHS Foundation Trust, Chertsey
  - 8260055 - NHS National Waiting Times Centre Golden Jubilee National Hospital, Clydebank
  - 8260058 - Royal Devon & Exeter NHS Foundation Trust, Exeter
  - 8260093 - The London North West Healthcare NHS Trust - Northwick Park, Harrow
  - 8260088 - Kettering General Hospital NHS Foundation Trust, Kettering
  - 8260043 - University Hospitals of Leicester NHS Trust - Glenfield, Leicester
  - 8260101 - United Lincolnshire Hospitals NHS Trust - Lincoln County Hospital, Lincoln
  - 8260086 - Manchester University NHS Foundation Trust - Manchester Royal Infirmary, Manchester
  - 8260065 - Milton Keynes Hospital NHS Foundation Trust, Milton Keynes
  - 8260134 - The Newcastle upon Tyne Hospitals NHS Foundation Trust - Fre, Newcastle upon Tyne
  - 8260068 - Morriston Hospital, Swansea
  - 8260066 - Torbay and South Devon NHS Foundation Trust - Torbay Hospital, Torquay
  - 8260099 - The Royal Wolverhampton NHS Trust - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson CM, Duffy D, Korjian S, Bahit MC, Chi G, Alexander JH, Lincoff AM, Heise M, Tricoci P, Deckelbaum LI, Mears SJ, Nicolau JC, Lopes RD, Merkely B, Lewis BS, Cornel JH, Trebacz J, Parkhomenko A, Libby P, Sacks FM, Povsic TJ, Bonaca M, Goodman SG, Bhatt DL, Tendera M, Steg PG, Ridker PM, Aylward P, Kastelein JJP, Bode C, Mahaffey KW, Nicholls SJ, Pocock SJ, Mehran R, Harrington RA; AEGIS-II Committees and Investigators. Apolipoprotein A1 Infusions and Cardiovascular Outcomes after Acute Myocardial Infarction. N Engl J Med. 2024 May 2;390(17):1560-1571. doi: 10.1056/NEJMoa2400969. Epub 2024 Apr 6. PMID 38587254
- [Background] Povsic TJ, Korjian S, Bahit MC, Chi G, Duffy D, Alexander JH, Vinereanu D, Tricoci P, Mears SJ, Deckelbaum LI, Bonaca M, Ridker PM, Goodman SG, Cornel JH, Lewis BS, Parkhomenko A, Lopes RD, Aylward P, Lincoff AM, Heise M, Sacks F, Nicolau JC, Merkely B, Trebacz J, Libby P, Nicholls SJ, Pocock S, Bhatt DL, Kastelein J, Bode C, Mahaffey KW, Steg PG, Tendera M, Bainey KR, Harrington RA, Mehran R, Duerschmied D, Kingwell BA, Gibson CM; AEGIS-II Committees and Investigators. Effect of Reconstituted Human Apolipoprotein A-I on Recurrent Ischemic Events in Survivors of Acute MI. J Am Coll Cardiol. 2024 Jun 4;83(22):2163-2174. doi: 10.1016/j.jacc.2024.03.396. Epub 2024 Apr 6. PMID 38588930
- [Derived] Gibson CM, Chi G, Duffy D, Bahit MC, White H, Korjian S, Alexander JH, Lincoff AM, Anschuetz G, Girgis IG, Nicolau JC, Lopes RD, Cornel JH, Bainey KR, Libby P, Sacks FM, Ridker PM, Goodman SG, Mahaffey KW, Nicholls SJ, Pocock SJ, Mehran R, Harrington RA; AEGIS-II Committees and Investigators. ApoA-I Infusions and Burden of Ischemic Events After Acute Myocardial Infarction: Insights From the AEGIS-II Trial. J Am Coll Cardiol. 2024 Nov 26;84(22):2185-2192. doi: 10.1016/j.jacc.2024.08.001. Epub 2024 Sep 2. PMID 39230545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 897 centers across 5 regions (North America, Latin America, Western Europe, Central and Eastern Europe, and Asia Pacific).
Pre-assignment Details: A total of 18,848 participants were screened, with 622 identified as screen failures. Of the screened participants, 18,226 were randomized in a 1:1 ratio to receive study interventions (CSL112 or Placebo).
Groups:
- CSL112: Participants received 6 grams of CSL112 (Apolipoprotein A-I [human] (apoA-I) purified from human plasma) once weekly via intravenous (IV) infusion for up to 4 weeks.
- Placebo: Participants received placebo (25% albumin solution diluted to 4.4%) once weekly via IV infusion for up to 4 weeks.
Period: Overall Study
Arm/Group | CSL112 | Placebo
Started | 9114 | 9112
Intent-to-treat (ITT) Analysis Set (The ITT analysis set comprised all randomized participants with the exception of 7 participants enrolled at site(s) excluded from analysis per sponsor decision.) | 9112 | 9107
Safety Analysis Set (SAS) (The SAS comprised all randomized participants in the ITT Analysis set who received any amount of the investigational product, and were analyzed based on the actual treatment received.) | 9010 | 9027
Completed | 9002 | 9020
Not Completed | 112 | 92
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 47 | 42
Not completed — Indirect contact | 32 | 29
Not completed — Other (Not specified) | 32 | 20

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the ITT analysis set. The ITT analysis set comprised all randomized participants with the exception of 7 participants enrolled at site(s) excluded from analysis per sponsor decision. The ITT analysis set utilized the treatment to which the participant was randomized regardless of the treatment actually received.
Groups:
- CSL112: Participants received 6 grams of CSL112 (apoA-I purified from human plasma) once weekly via IV infusion for up to 4 weeks.
- Total: Total of all reporting groups
Arm/Group | CSL112 | Placebo | Total
Number analyzed (Participants) | 9112 | 9107 | 18219
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (10.09) | 65.4 (10.21) | 65.5 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2326 | 2386 | 4712
  Male | 6786 | 6721 | 13507
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1566 | 1596 | 3162
  Not Hispanic or Latino | 7410 | 7383 | 14793
  Unknown or Not Reported | 136 | 128 | 264
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 51 | 36 | 87
  Asian | 743 | 781 | 1524
  Black or African American | 181 | 181 | 362
  Native Hawaiian or other Pacific Islander | 8 | 10 | 18
  White | 7769 | 7698 | 15467
  Multiracial or other | 314 | 356 | 670
  Not Reported by subject | 46 | 45 | 91

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of Any Component of Composite MACE (CV Death, MI, or Stroke)
Description: MACE (Major adverse cardiovascular event[s])(CV [cardiovascular] death, MI [Myocardial Infarction], or stroke).
Time Frame: From the time of randomization through 90 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 9112 | 9107
Participants | 439 | 472
Statistical Analysis 1: Comparison: CSL112 vs Placebo; Test type: Superiority; p = 0.121, Cox proportional hazards regression — 1-sided p-value; Hazard Ratio (HR) = 0.925, 95% CI 2-sided [0.8126 to 1.0538]

2. Secondary Outcome: Total Number of Hospitalizations for Coronary, Cerebral, and Peripheral Ischemia
Description: The total number of hospitalizations and individual hospitalizations due to coronary, cerebral, and peripheral ischemia were reported.
Time Frame: From the time of randomization through 90 days
Population: as for baseline characteristics
Measure: Number; unit: hospitalizations
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 9112 | 9107
hospitalizations
  Total hospitalizations | 433 | 442
  Coronary ischemia | 367 | 376
  Cerebral ischemia | 39 | 36
  Peripheral ischemia | 27 | 30
Statistical Analysis 1: Comparison: CSL112 vs Placebo; Test type: Superiority; p = 0.341, Negative binomial regression model — 1-sided p-value; Rate ratio = 0.971, 95% CI 2-sided [0.8442 to 1.1171]

3. Secondary Outcome: Number of Participants With First Occurrence of CV Death, MI, or Stroke
Time Frame: From the time of randomization through 180 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 9112 | 9107
Participants | 622 | 683
Statistical Analysis 1: Comparison: CSL112 vs Placebo; Test type: Superiority; p = 0.038, Cox proportional hazards regression — 1-sided p-value; Hazard Ratio (HR) = 0.907, 95% CI 2-sided [0.8132 to 1.0106]

4. Secondary Outcome: Number of Participants With First Occurrence of CV Death, MI, or Stroke
Time Frame: From the time of randomization through 365 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 9112 | 9107
Participants | 885 | 944
Statistical Analysis 1: Comparison: CSL112 vs Placebo; Test type: Superiority; p = 0.069, Cox proportional hazards regression — 1-sided p-value; Hazard Ratio (HR) = 0.933, 95% CI 2-sided [0.8511 to 1.0224]

5. Secondary Outcome: Number of Participants With Occurrence of CV Death
Time Frame: From the time of randomization through 90 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 9112 | 9107
Participants | 107 | 128
Statistical Analysis 1: Comparison: CSL112 vs Placebo; Test type: Superiority; p = 0.074, Cox proportional hazards regression — 1-sided p-value; Hazard Ratio (HR) = 0.827, 95% CI 2-sided [0.6399 to 1.0695]

6. Secondary Outcome: Number of Participants With First Occurrence of MI
Time Frame: From the time of randomization through 90 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 9112 | 9107
Participants | 312 | 342
Statistical Analysis 1: Comparison: CSL112 vs Placebo; Test type: Superiority; p = 0.113, Cox proportional hazards regression — 1-sided p-value; Hazard Ratio (HR) = 0.909, 95% CI 2-sided [0.7801 to 1.0603]

7. Secondary Outcome: Number of Participants With First Occurrence of Stroke
Time Frame: From the time of randomization through 90 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 9112 | 9107
Participants | 57 | 49
Statistical Analysis 1: Comparison: CSL112 vs Placebo; Test type: Superiority; p = 0.767, Cox proportional hazards regression — 1-sided p-value; Hazard Ratio (HR) = 1.153, 95% CI 2-sided [0.7867 to 1.6886]

8. Secondary Outcome: Number of Participants With First Occurrence of CV Death, Type 1 MI or Stroke
Time Frame: From the time of randomization through 90, 180 and 365 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 9112 | 9107
Participants
  Through Day 90 | 272 | 308
  Through Day 180 | 400 | 444
  Through Day 365 | 594 | 639

9. Secondary Outcome: Number of Participants With Occurrence of All-cause Death
Time Frame: From the time of randomization through 365 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 9112 | 9107
Participants | 341 | 345

10. Secondary Outcome: Number of Participants With Adverse Events
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal, clinically significant laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product.
Time Frame: From the start of treatment through 90 days
Population: Analysis was performed on the Safety analysis set (SAS). The SAS comprised all participants in the ITT Analysis set who received any amount of the investigational product, and were analyzed based on the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 9010 | 9027
Participants | 3938 | 3927

11. Secondary Outcome: Percentage of Participants With Adverse Events
Description: as for outcome 10
Time Frame: From the start of treatment through 90 days
Population: Analysis was performed on the SAS. The SAS comprised all participants in the ITT Analysis set who received any amount of the investigational product, and were analyzed based on the actual treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 9010 | 9027
percentage of participants | 43.7 | 43.5

12. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Description: Treatment-related AEs were AEs considered by the Investigator to have a causal relationship to the investigational product.
Time Frame: From the start of treatment through 379 days (Day 365 + 14 days of follow up)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 9010 | 9027
Participants | 350 | 304

13. Secondary Outcome: Percentage of Participants With Treatment-related Adverse Events
Description: Treatment-related AEs were AEs considered by the Investigator to have a causal relationship to the investigational product. As per the study statistical analysis plan (SAP), descriptive percentages were displayed to one decimal place, hence the percentage values were rounded off and presented.
Time Frame: From the start of treatment through 379 days (Day 365 + 14 days of follow up)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 9010 | 9027
percentage of participants | 3.9 | 3.4

14. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: SAE was defined as any untoward medical occurrence that at any dose: results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is a medically significant event.
Time Frame: From the start of treatment through 379 days (Day 365 + 14 days of follow up)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 9010 | 9027
Participants | 1514 | 1557

15. Secondary Outcome: Percentage of Participants With SAEs
Description: SAE was defined as any untoward medical occurrence that at any dose: results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect or is a medically significant event. As per the study SAP, descriptive percentages were displayed to one decimal place, hence the percentage values were rounded off and presented.
Time Frame: From the start of treatment through 379 days (Day 365 + 14 days of follow up)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 9010 | 9027
percentage of participants | 16.8 | 17.2

16. Secondary Outcome: Number of Participants With a Shift From Baseline to Worst Post-treatment Value in Clinical Laboratory Assessments
Description: Clinical laboratory assessments included assessment of Hematology (hemoglobin, hematocrit, leukocytes and platelets) and Biochemistry (alkaline phosphatase [ALP], alanine aminotransferase [ALT], aspartate aminotransferase [AST], bilirubin, direct bilirubin, indirect bilirubin and estimated glomerular filtration rate [eGFR]). The number of participants with a shift from the Baseline value to the worst post-treatment value (low, normal, or high) was reported. The worst criterion for the parameters is as follows: hematocrit - low, hemoglobin - low, leukocytes - high, platelets - low, ALT - high, ALP - high, AST - high, bilirubin - high, direct bilirubin - high, indirect bilirubin - high, eGFR - severe impairment.
Time Frame: Baseline and 29 days
Population: Analysis was performed on the SAS. The SAS comprised all participants in the ITT Analysis set who received any amount of the investigational product, and were analyzed based on the actual treatment received. Here, the Overall Number of Participants Analyzed (N), included all participants who were evaluated for this outcome measure and the Number Analyzed (n), included all participants who were evaluated for this outcome measure for the specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 8372 | 8392
Participants
  Hematocrit - High to Low: number analyzed (Participants) | 6848 | 6810
  Hematocrit - High to Low | 0 | 1
  Hematocrit - Normal to Low: number analyzed (Participants) | 6848 | 6810
  Hematocrit - Normal to Low | 365 | 393
  Hemoglobin - High to Low: number analyzed (Participants) | 7235 | 7185
  Hemoglobin - High to Low | 0 | 1
  Hemoglobin - Normal to Low: number analyzed (Participants) | 7235 | 7185
  Hemoglobin - Normal to Low | 457 | 447
  Leukocytes - Normal to High: number analyzed (Participants) | 7229 | 7184
  Leukocytes - Normal to High | 267 | 271
  Leukocytes - Low to High: number analyzed (Participants) | 7229 | 7184
  Leukocytes - Low to High | 2 | 1
  Platelets - High to Low: number analyzed (Participants) | 7138 | 7064
  Platelets - High to Low | 0 | 0
  Platelets - Normal to Low: number analyzed (Participants) | 7138 | 7064
  Platelets - Normal to Low | 92 | 114
  ALT - Normal to High: number analyzed (Participants) | 7904 | 7949
  ALT - Normal to High | 658 | 612
  ALT - Low to High: number analyzed (Participants) | 7904 | 7949
  ALT - Low to High | 0 | 0
  ALP - Normal to High: number analyzed (Participants) | 8341 | 8366
  ALP - Normal to High | 307 | 350
  ALP - Low to High: number analyzed (Participants) | 8341 | 8366
  ALP - Low to High | 1 | 0
  AST - Normal to High: number analyzed (Participants) | 7910 | 7911
  AST - Normal to High | 239 | 253
  AST - Low to High: number analyzed (Participants) | 7910 | 7911
  AST - Low to High | 2 | 0
  Bilirubin - Normal to High: number analyzed (Participants) | 8281 | 8284
  Bilirubin - Normal to High | 73 | 112
  Bilirubin - Low to High: number analyzed (Participants) | 8281 | 8284
  Bilirubin - Low to High | 0 | 1
  Direct Bilirubin - Normal to High: number analyzed (Participants) | 7273 | 7317
  Direct Bilirubin - Normal to High | 18 | 21
  Direct Bilirubin - Low to High: number analyzed (Participants) | 7273 | 7317
  Direct Bilirubin - Low to High | 0 | 0
  Indirect Bilirubin - Normal to High: number analyzed (Participants) | 7269 | 7309
  Indirect Bilirubin - Normal to High | 31 | 42
  Indirect Bilirubin - Low to High: number analyzed (Participants) | 7269 | 7309
  Indirect Bilirubin - Low to High | 0 | 0
  eGFR - Normal to Severe Impairment | 1 | 2
  eGFR - Mild Impairment to Severe Impairment | 15 | 9
  eGFR - Moderate Impairment to Severe Impairment | 91 | 99

17. Secondary Outcome: Percentage of Participants With a Shift From Baseline to Worst Post-treatment Value in Clinical Laboratory Assessments
Description: Clinical laboratory assessments included assessment of Hematology (hemoglobin, hematocrit, leukocytes and platelets) and Biochemistry (ALP, ALT, AST, bilirubin, direct bilirubin, indirect bilirubin and eGFR). Percentage of participants with a shift from the Baseline value to the worst post-treatment value (low, normal, or high) was reported. The worst criterion for the parameters is as follows: hematocrit - low, hemoglobin - low, leukocytes - high, platelets - low, ALT - high, ALP - high, AST - high, bilirubin - high, direct bilirubin - high, indirect bilirubin - high, eGFR - severe impairment. As per the study SAP, descriptive percentages were displayed to one decimal place, hence the percentage values were rounded off and presented.
Time Frame: Baseline and 29 days
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 8372 | 8392
percentage of participants
  Hematocrit - High to Low: number analyzed (Participants) | 6848 | 6810
  Hematocrit - High to Low | 0.0 | 0.0
  Hematocrit - Normal to Low: number analyzed (Participants) | 6848 | 6810
  Hematocrit - Normal to Low | 5.3 | 5.8
  Hemoglobin - High to Low: number analyzed (Participants) | 7235 | 7185
  Hemoglobin - High to Low | 0.0 | 0.0
  Hemoglobin - Normal to Low: number analyzed (Participants) | 7235 | 7185
  Hemoglobin - Normal to Low | 6.3 | 6.2
  Leukocytes - Normal to High: number analyzed (Participants) | 7229 | 7184
  Leukocytes - Normal to High | 3.7 | 3.8
  Leukocytes - Low to High: number analyzed (Participants) | 7229 | 7184
  Leukocytes - Low to High | 0.0 | 0.0
  Platelets - High to Low: number analyzed (Participants) | 7138 | 7064
  Platelets - High to Low | 0.0 | 0.0
  Platelets - Normal to Low: number analyzed (Participants) | 7138 | 7064
  Platelets - Normal to Low | 1.3 | 1.6
  ALT - Normal to High: number analyzed (Participants) | 7904 | 7949
  ALT - Normal to High | 8.3 | 7.7
  ALT - Low to High: number analyzed (Participants) | 7904 | 7949
  ALT - Low to High | 0.0 | 0.0
  ALP - Normal to High: number analyzed (Participants) | 8341 | 8366
  ALP - Normal to High | 3.7 | 4.2
  ALP - Low to High: number analyzed (Participants) | 8341 | 8366
  ALP - Low to High | 0.0 | 0.0
  AST - Normal to High: number analyzed (Participants) | 7910 | 7911
  AST - Normal to High | 3.0 | 3.2
  AST - Low to High: number analyzed (Participants) | 7910 | 7911
  AST - Low to High | 0.0 | 0.0
  Bilirubin - Normal to High: number analyzed (Participants) | 8281 | 8284
  Bilirubin - Normal to High | 0.9 | 1.4
  Bilirubin - Low to High: number analyzed (Participants) | 8281 | 8284
  Bilirubin - Low to High | 0.0 | 0.0
  Direct Bilirubin - Normal to High: number analyzed (Participants) | 7273 | 7317
  Direct Bilirubin - Normal to High | 0.2 | 0.3
  Direct Bilirubin - Low to High: number analyzed (Participants) | 7273 | 7317
  Direct Bilirubin - Low to High | 0.0 | 0.0
  Indirect Bilirubin - Normal to High: number analyzed (Participants) | 7269 | 7309
  Indirect Bilirubin - Normal to High | 0.4 | 0.6
  Indirect Bilirubin - Low to High: number analyzed (Participants) | 7269 | 7309
  Indirect Bilirubin - Low to High | 0.0 | 0.0
  eGFR - Normal to Severe Impairment | 0.0 | 0.0
  eGFR - Mild Impairment to Severe Impairment | 0.2 | 0.1
  eGFR - Moderate Impairment to Severe Impairment | 1.1 | 1.2

18. Secondary Outcome: Change From Baseline in Hematology Parameters
Description: Hematology parameters included Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets.
Time Frame: From Baseline to Day 29
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 7073 | 7021
10^9 cells per liter
  Basophils: number analyzed (Participants) | 7061 | 7011
  Basophils | 0.004 (0.0455) | 0.005 (0.0462)
  Eosinophils: number analyzed (Participants) | 7061 | 7011
  Eosinophils | 0.045 (0.1766) | 0.047 (0.1727)
  Leukocytes | -1.024 (2.2905) | -0.969 (2.2683)
  Lymphocytes: number analyzed (Participants) | 7061 | 7011
  Lymphocytes | 0.084 (0.5534) | 0.080 (0.5409)
  Monocytes: number analyzed (Participants) | 7061 | 7011
  Monocytes | -0.089 (0.1886) | -0.087 (0.1961)
  Neutrophils: number analyzed (Participants) | 7061 | 7011
  Neutrophils | -1.068 (2.0892) | -1.011 (2.0343)
  Platelets: number analyzed (Participants) | 6985 | 6908
  Platelets | 0.4 (56.09) | -1.4 (55.31)

19. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Time Frame: From Baseline to Day 29
Population: Analysis was performed on the SAS. The SAS comprised all participants in the ITT Analysis set who received any amount of the investigational product, and were analyzed based on the actual treatment received. Here, the Overall Number of Participants Analyzed (N), included all participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: liter per liter (L/L)
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 6698 | 6651
liter per liter (L/L) | -0.003 (0.0382) | -0.004 (0.0381)

20. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin
Time Frame: From Baseline to Day 29
Population: Analysis was performed on the SAS. The SAS comprised all participants in the ITT Analysis set who received any amount of the investigational product, and were analyzed based on the actual treatment received. Here, Overall Number of Participants Analyzed (N), included all participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 7074 | 7021
grams per liter (g/L) | -1.1 (11.96) | -1.3 (12.08)

21. Secondary Outcome: Change From Baseline in Hepatic Parameters
Description: Hepatic parameters included ALT, ALP and AST.
Time Frame: From Baseline to Day 29
Population: Analysis was performed on the SAS. The SAS comprised all participants in the ITT Analysis set who received any amount of the investigational product, and were analyzed based on the actual treatment received. Here, the Overall Number of Participants Analyzed (N), included all participants who were evaluated for this outcome measure and the Number Analyzed (n), included all participants who were evaluated for this outcome measure for each specified category.
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 8079 | 8072
units per liter
  ALT: number analyzed (Participants) | 7628 | 7630
  ALT | -5.5 (25.52) | -6.5 (28.91)
  ALP | 3.2 (26.13) | 4.5 (24.55)
  AST: number analyzed (Participants) | 7616 | 7574
  AST | -21.2 (41.90) | -20.7 (61.63)

22. Secondary Outcome: Change From Baseline in Hepatic Parameter: Bilirubin
Time Frame: From Baseline to Day 29
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: micromol per liter (umol/L)
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 8005 | 7983
micromol per liter (umol/L)
  Bilirubin | -2.6 (4.71) | -1.9 (5.05)
  Direct Bilirubin: number analyzed (Participants) | 6961 | 6958
  Direct Bilirubin | -0.4 (1.32) | -0.3 (1.75)
  Indirect Bilirubin: number analyzed (Participants) | 6957 | 6950
  Indirect Bilirubin | -2.0 (3.85) | -1.4 (3.90)

23. Secondary Outcome: Change From Baseline in Renal Parameter: Serum Creatinine
Time Frame: From Baseline to Day 29
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 8114 | 8101
umol/L | 2.4 (24.39) | 2.1 (21.23)

24. Secondary Outcome: Change From Baseline in Renal Parameter: eGFR
Time Frame: From Baseline to Day 29
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: milliliter per minute per 1.73 meter^2
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 8112 | 8098
milliliter per minute per 1.73 meter^2 | -1.3 (11.87) | -1.2 (12.15)

25. Secondary Outcome: Change From Baseline in Renal Parameter: Blood Urea Nitrogen
Time Frame: From Baseline to Day 29
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: millimoles per liter
Arm/Group | CSL112 | Placebo
Number analyzed (Participants) | 8114 | 8105
millimoles per liter | 0.0 (2.76) | 0.0 (2.67)

ADVERSE EVENTS:
Time Frame: All AEs were collected through Day 90 and AEs related to study drug, those leading to its discontinuation, withdrawal of consent, all-cause mortality, Other AEs and all SAEs were collected up to Day 379 (Day 365+ 14 days of follow-up)
Description: All-cause mortality was monitored/assessed for the ITT population, but Serious and Other AEs were only monitored/assessed for the SAS population. The SAS included all ITT participants (with the exception of participants enrolled at site(s) excluded from analysis due to concerns regarding data integrity) who received any investigational product and analyzed based on actual treatment received. The SAS was the primary population for summarizing and reporting safety data (SAEs and Other AEs).
Arm/Group | CSL112 | Placebo
All-Cause Mortality (participants affected / at risk) | 348/9112 | 355/9107
Serious Adverse Events (participants affected / at risk) | 1514/9010 | 1557/9027
Other Adverse Events (participants affected / at risk) | 0/9010 | 0/9027
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL112 (N=9010) | Placebo (N=9027)
Angina pectoris (Cardiac disorders) | 106 (107) | 84 (89)
Angina unstable (Cardiac disorders) | 69 (73) | 59 (63)
Cardiac failure (Cardiac disorders) | 54 (61) | 64 (67)
Atrial fibrillation (Cardiac disorders) | 48 (50) | 48 (53)
Coronary artery disease (Cardiac disorders) | 23 (23) | 27 (28)
Ventricular tachycardia (Cardiac disorders) | 20 (21) | 21 (24)
Acute myocardial infarction (Cardiac disorders) | 19 (19) | 29 (29)
Myocardial infarction (Cardiac disorders) | 14 (15) | 16 (16)
Myocardial ischaemia (Cardiac disorders) | 14 (15) | 19 (19)
Cardiac failure congestive (Cardiac disorders) | 14 (14) | 23 (24)
Atrial flutter (Cardiac disorders) | 12 (12) | 15 (16)
Cardiac arrest (Cardiac disorders) | 11 (11) | 13 (13)
Pericarditis (Cardiac disorders) | 10 (11) | 6 (6)
Cardiogenic shock (Cardiac disorders) | 10 (10) | 6 (6)
Coronary artery stenosis (Cardiac disorders) | 9 (9) | 7 (7)
Acute coronary syndrome (Cardiac disorders) | 8 (8) | 6 (6)
Atrioventricular block complete (Cardiac disorders) | 8 (8) | 10 (11)
Sinus node dysfunction (Cardiac disorders) | 8 (8) | 8 (8)
Cardiac failure acute (Cardiac disorders) | 7 (8) | 12 (12)
Left ventricular failure (Cardiac disorders) | 7 (8) | 5 (5)
Supraventricular tachycardia (Cardiac disorders) | 7 (8) | 4 (4)
Bradycardia (Cardiac disorders) | 7 (7) | 8 (8)
Atrioventricular block second degree (Cardiac disorders) | 5 (5) | 5 (5)
Ischaemic cardiomyopathy (Cardiac disorders) | 5 (5) | 4 (4)
Mitral valve incompetence (Cardiac disorders) | 5 (5) | 4 (4)
Ventricular fibrillation (Cardiac disorders) | 5 (5) | 6 (6)
Torsade de pointes (Cardiac disorders) | 4 (6) | 2 (2)
Atrioventricular block (Cardiac disorders) | 4 (4) | 7 (7)
Coronary artery occlusion (Cardiac disorders) | 4 (4) | 5 (5)
Dressler's syndrome (Cardiac disorders) | 4 (4) | 6 (7)
Pericardial effusion (Cardiac disorders) | 4 (4) | 5 (5)
Postinfarction angina (Cardiac disorders) | 4 (4) | 6 (6)
Ventricular extrasystoles (Cardiac disorders) | 4 (4) | 3 (5)
Cardio-respiratory arrest (Cardiac disorders) | 3 (6) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 3 (3) | 4 (4)
Coronary artery perforation (Cardiac disorders) | 3 (3) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 3 (3)
Arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac ventricular thrombosis (Cardiac disorders) | 2 (2) | 5 (5)
Mitral valve stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial injury (Cardiac disorders) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 5 (7)
Sinus arrest (Cardiac disorders) | 2 (2) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac asthma (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac discomfort (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Chronic coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 4 (4)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 2 (2)
Low cardiac output syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial rupture (Cardiac disorders) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 3 (3)
Anginal equivalent (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 2 (2)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 3 (3)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial mass (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Trifascicular block (Cardiac disorders) | 0 (0) | 1 (1)
Ventricle rupture (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 97 (99) | 89 (93)
COVID-19 pneumonia (Infections and infestations) | 52 (52) | 46 (47)
COVID-19 (Infections and infestations) | 42 (42) | 48 (49)
Urinary tract infection (Infections and infestations) | 37 (38) | 36 (39)
Sepsis (Infections and infestations) | 26 (26) | 26 (26)
Urosepsis (Infections and infestations) | 12 (13) | 8 (8)
Gastroenteritis (Infections and infestations) | 12 (12) | 7 (7)
Cellulitis (Infections and infestations) | 9 (9) | 17 (19)
Bronchitis (Infections and infestations) | 7 (7) | 6 (6)
Respiratory tract infection (Infections and infestations) | 7 (7) | 2 (2)
Septic shock (Infections and infestations) | 7 (7) | 23 (23)
Osteomyelitis (Infections and infestations) | 6 (6) | 7 (9)
Influenza (Infections and infestations) | 5 (5) | 7 (7)
Peritonitis (Infections and infestations) | 5 (5) | 0 (0)
Postoperative wound infection (Infections and infestations) | 5 (5) | 4 (4)
Pyelonephritis (Infections and infestations) | 5 (5) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 4 (4)
Appendicitis (Infections and infestations) | 4 (5) | 6 (6)
Pneumonia bacterial (Infections and infestations) | 4 (4) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (4) | 7 (8)
Bacteraemia (Infections and infestations) | 3 (3) | 1 (1)
Endocarditis (Infections and infestations) | 3 (3) | 3 (3)
Staphylococcal bacteraemia (Infections and infestations) | 3 (3) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 2 (3) | 2 (2)
Pneumonia aspiration (Infections and infestations) | 2 (3) | 6 (6)
Abscess limb (Infections and infestations) | 2 (2) | 2 (2)
Cholecystitis infective (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 3 (3)
Epididymitis (Infections and infestations) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 4 (4)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 2 (2)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Intervertebral discitis (Infections and infestations) | 2 (2) | 2 (5)
Localised infection (Infections and infestations) | 2 (2) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 2 (2) | 1 (1)
Parapharyngeal space infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 2 (2)
Viral infection (Infections and infestations) | 2 (2) | 1 (1)
Lung abscess (Infections and infestations) | 1 (2) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 3 (3)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Aortitis syphilitic (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 2 (2)
Arthritis infective (Infections and infestations) | 1 (1) | 1 (1)
Babesiosis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Chikungunya virus infection (Infections and infestations) | 1 (1) | 0 (0)
Complicated appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Coronavirus pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 2 (2)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 1 (1) | 0 (0)
Emphysematous cystitis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 2 (2)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Groin infection (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis E (Infections and infestations) | 1 (1) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 1 (1) | 1 (1)
Medical device site infection (Infections and infestations) | 1 (1) | 2 (2)
Medical device site joint infection (Infections and infestations) | 1 (1) | 0 (0)
Muscle abscess (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Salmonella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Sternitis (Infections and infestations) | 1 (1) | 0 (0)
Thrombophlebitis septic (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Vascular access site infection (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 2 (3)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Bacterial prostatitis (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Citrobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 2 (2)
Cystitis klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Erysipelothrix sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 2 (2)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Gas gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 3 (3)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 2 (2)
Otitis externa (Infections and infestations) | 0 (0) | 2 (2)
Peritoneal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia acinetobacter (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 1 (1)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1)
Pyonephrosis (Infections and infestations) | 0 (0) | 1 (1)
Pyuria (Infections and infestations) | 0 (0) | 2 (2)
Retroperitoneal abscess (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 2 (2)
Strongyloidiasis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 (14) | 19 (19)
Gastritis (Gastrointestinal disorders) | 10 (10) | 7 (10)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 8 (10)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 7 (8) | 3 (4)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 (7) | 3 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 (7) | 4 (5)
Rectal haemorrhage (Gastrointestinal disorders) | 6 (8) | 5 (5)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 6 (6) | 7 (7)
Pancreatitis acute (Gastrointestinal disorders) | 6 (6) | 12 (15)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 5 (5)
Melaena (Gastrointestinal disorders) | 5 (5) | 6 (7)
Colitis ischaemic (Gastrointestinal disorders) | 4 (4) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 8 (8)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 4 (4) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 4 (4) | 5 (5)
Duodenal ulcer (Gastrointestinal disorders) | 3 (3) | 5 (5)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (3) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 4 (4)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gingival bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 2 (2) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (5)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (2)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Heyde's syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (2)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal erosion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 4 (4)
Pancreatic atrophy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis relapsing (Gastrointestinal disorders) | 0 (0) | 2 (2)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 2 (2)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 6 (9)
Acute kidney injury (Renal and urinary disorders) | 68 (72) | 66 (71)
Renal impairment (Renal and urinary disorders) | 15 (15) | 14 (17)
Haematuria (Renal and urinary disorders) | 14 (16) | 10 (14)
Renal failure (Renal and urinary disorders) | 12 (13) | 14 (14)
Nephropathy toxic (Renal and urinary disorders) | 11 (11) | 6 (6)
Urinary retention (Renal and urinary disorders) | 10 (10) | 6 (6)
Nephrolithiasis (Renal and urinary disorders) | 6 (6) | 8 (8)
Chronic kidney disease (Renal and urinary disorders) | 4 (4) | 4 (4)
Ureterolithiasis (Renal and urinary disorders) | 4 (4) | 2 (2)
Calculus urinary (Renal and urinary disorders) | 3 (4) | 1 (2)
Renal colic (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Bladder disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1)
Pyelocaliectasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral haemorrhage (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder diverticulum (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 2 (2)
Calculus urethral (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis erosive (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 2 (3)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (2)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal salt-wasting syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Vesical fistula (Renal and urinary disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 92 (97) | 78 (99)
Pyrexia (General disorders) | 12 (12) | 8 (9)
Chest pain (General disorders) | 7 (7) | 15 (15)
Vascular stent stenosis (General disorders) | 7 (7) | 6 (6)
General physical health deterioration (General disorders) | 5 (6) | 1 (1)
Gait disturbance (General disorders) | 4 (4) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 2 (2)
Medical device site haematoma (General disorders) | 1 (1) | 1 (1)
Death (General disorders) | 1 (1) | 2 (2)
Drowning (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 1 (1)
Infusion site reaction (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Vascular stent occlusion (General disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 10 (10)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Drug intolerance (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (3)
Hernia (General disorders) | 0 (0) | 1 (1)
Immune-mediated polyserositis (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2)
Medical device site haemorrhage (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Physical deconditioning (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 2 (2)
Vascular stent thrombosis (General disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 21 (28) | 29 (41)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 13 (14)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 12 (12)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (8)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 11 (13)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (8)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Diaphragmatic abnormal relaxation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 7 (7)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 7 (8)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (5)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Lung squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Paget's disease of nipple (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urethral cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Borderline mucinous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ciliary body melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypopharyngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell cancer of renal pelvis and ureter metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 11 (11) | 11 (11)
Subdural haematoma (Injury, poisoning and procedural complications) | 9 (9) | 6 (7)
Femur fracture (Injury, poisoning and procedural complications) | 8 (8) | 11 (11)
Head injury (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)
Hip fracture (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 5 (5) | 7 (7)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Rib fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Craniofacial fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 2 (2) | 1 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Pancreatic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chemical burns of eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Costal cartilage fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eschar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exposure to SARS-CoV-2 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Renal transplant failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic renal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Gas poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal anastomotic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyphaema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication circulatory (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Radiation proctitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Respiratory tract procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access site dissection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 17 (19) | 15 (15)
Aortic aneurysm (Vascular disorders) | 11 (11) | 4 (4)
Hypertension (Vascular disorders) | 11 (11) | 14 (15)
Hypertensive crisis (Vascular disorders) | 10 (10) | 12 (15)
Deep vein thrombosis (Vascular disorders) | 7 (7) | 3 (3)
Peripheral arterial occlusive disease (Vascular disorders) | 7 (7) | 11 (11)
Aortic stenosis (Vascular disorders) | 4 (4) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 7 (7)
Peripheral ischaemia (Vascular disorders) | 4 (4) | 5 (5)
Haematoma (Vascular disorders) | 3 (3) | 3 (3)
Aortic dissection (Vascular disorders) | 2 (2) | 0 (0)
Hypertensive emergency (Vascular disorders) | 2 (2) | 3 (3)
Phlebitis (Vascular disorders) | 2 (2) | 5 (5)
Thrombophlebitis (Vascular disorders) | 2 (2) | 3 (3)
Angiodysplasia (Vascular disorders) | 1 (1) | 1 (1)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Dialysis hypotension (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 2 (2)
Granulomatosis with polyangiitis (Vascular disorders) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive urgency (Vascular disorders) | 1 (1) | 3 (3)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 5 (5)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 1 (1)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Arterial rupture (Vascular disorders) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 3 (3)
Leriche syndrome (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 3 (3)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 23 (24) | 26 (26)
Transient ischaemic attack (Nervous system disorders) | 6 (6) | 10 (10)
Carotid artery stenosis (Nervous system disorders) | 5 (5) | 5 (5)
Dizziness (Nervous system disorders) | 5 (5) | 5 (5)
Loss of consciousness (Nervous system disorders) | 5 (5) | 0 (0)
Seizure (Nervous system disorders) | 5 (5) | 4 (4)
Presyncope (Nervous system disorders) | 4 (4) | 10 (10)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 4 (4)
Epilepsy (Nervous system disorders) | 3 (3) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 3 (3) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (3) | 1 (2)
Cerebrovascular disorder (Nervous system disorders) | 2 (2) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 4 (4)
Neuralgia (Nervous system disorders) | 1 (2) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (2) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (2) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Carotid sinus syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 4 (4)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 1 (2)
Diabetic coma (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhage intracranial (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 1 (1) | 0 (0)
Post stroke epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Pseudoradicular syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 1 (2)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 2 (2)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 12 (14) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (10) | 14 (14)
Dehydration (Metabolism and nutrition disorders) | 9 (9) | 6 (6)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 7 (7) | 6 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 9 (9)
Gout (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Failure to thrive (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 40 (45) | 39 (43)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 9 (9) | 8 (9)
Blood loss anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acquired haemophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 57 (64) | 12 (13)
Cholecystitis acute (Hepatobiliary disorders) | 11 (11) | 17 (18)
Liver injury (Hepatobiliary disorders) | 7 (7) | 12 (12)
Cholelithiasis (Hepatobiliary disorders) | 6 (6) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 4 (4) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 2 (2) | 2 (2)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic fibrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 4 (4)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 15 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Costochondritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 5 (5) | 1 (1)
Hepatic enzyme increased (Investigations) | 4 (4) | 1 (1)
Liver function test abnormal (Investigations) | 3 (3) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Ejection fraction decreased (Investigations) | 2 (2) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2) | 5 (5)
Influenza A virus test positive (Investigations) | 2 (2) | 0 (0)
Anticoagulation drug level abnormal (Investigations) | 1 (1) | 1 (1)
Bacterial test positive (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Inflammatory marker increased (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 2 (2)
Troponin I increased (Investigations) | 1 (1) | 0 (0)
Angiogram peripheral abnormal (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 2 (3)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Gram stain positive (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Pulmonary arterial pressure increased (Investigations) | 0 (0) | 1 (1)
Staphylococcus test positive (Investigations) | 0 (0) | 1 (1)
Troponin T increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 8 (8) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Necrotic angiodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic wound (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 6 (6)
Panic attack (Psychiatric disorders) | 2 (2) | 2 (2)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Tobacco withdrawal symptoms (Psychiatric disorders) | 1 (1) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 4 (4)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 2 (3)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 5 (5) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 4 (5) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Cytokine storm (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 2 (2)
Vertigo positional (Ear and labyrinth disorders) | 4 (4) | 3 (3)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 4 (4)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0)
Eye allergy (Eye disorders) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Retinopathy hypertensive (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Purtscher retinopathy (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Tolosa-Hunt syndrome (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 2 (2)
Prostatitis (Reproductive system and breast disorders) | 3 (3) | 4 (4)
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 (3) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatic disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypoaldosteronism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Adrenocortical insufficiency acute (Endocrine disorders) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 1 (2) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Loss of personal independence in daily activities (Social circumstances) | 1 (1) | 2 (2)
Victim of abuse (Social circumstances) | 1 (1) | 0 (0)
Physical disability (Social circumstances) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Lymphatic malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Assisted suicide (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT03473223/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT03473223/SAP_001.pdf